Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – Tofacitinib vs Abatacept

NCT04529876

November 24, 2020

### 1. Comparison Details

### a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>tofacitinib versus abatacept</u> for rheumatoid arthritis.

### b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

### 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

## 3. Data Source(s)

Medicare, 2007-2017

### 4. Study Design Diagrams





#### 5. Cohort Identification

### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing to facitinib to abatacept. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of to facitinib or abatacept (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

### b. Key details regarding cohort creation

#### Index date:

Day of initiation of new tofacitinib or abatacept use

### Inclusion criteria for analyses 1, 3, 4:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of tofacitinib or abatacept any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least one inpatient or one outpatient claim with rheumatoid arthritis diagnosis recorded in 365 days prior to and including index date
- No history of nursing home admission recorded in 365 days prior to and including index date

### Inclusion criteria for analysis 2:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of tofacitinib or abatacept any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least one inpatient or one outpatient claim with rheumatoid arthritis diagnosis recorded in 365 days prior to and including index date
- 180-day continuous use of tofacitinib or abatacept starting on the index date
- No history of nursing home admission recorded in 365 days prior to and including index date

# c. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 7,964,044 |
| Did not meet cohort entry criteria | -7,886,909 | 77,135 |
| Excluded due to insufficient enrollment | -30,469 | 46,666 |
| Excluded due to prior use of referent | -13,278 | 33,388 |
| Excluded due to prior use of exposure | -1,820 | 31,568 |
| Excluded because patient qualified in >1 exposure category | 0 | 31,568 |
| Excluded based on Dementia Exclusion | -323 | 31,245 |
| Excluded based on RA Diagnosis | -74 | 31,171 |
| Excluded based on Nursing Home Admission | -155 | 31,016 |
| Excluded because patient did not begin follow-up | -1,552 | 29,464 |
| Patients in tofacitinib group | | 4,456 |
| Patients in abatacept group | | 25,008 |
| Final cohort | | 29,464 |

## 6. Variables

# a. Exposure-related variables:

Study drug:

The study exposure of interest is initiation of tofacitinib

Comparator:

Initiators of tofacitinib will be compared to initiators of Abatacept

## b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|---------------------------------------|------------------|
| Diabetes Depression | |
| Obesity | Anxiety |
| Hypertension | Bipolar disorder |
| Coronary artery disease Schizophrenia | |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of hospitalizations |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of rheumatologist visits |
| Pneumococcal vaccination | Number of C-reactive protein tests ordered |
| Herpes zoster vaccination | Osteoporosis |

| Bone mineral density test | Fractures |
|-----------------------------------|----------------------------|
| Number of distinct generic agents | Falls |
| Number of emergency room visits | Use of supplemental oxygen |
| Number of outpatient visits | Combined comorbidity score |

| Comedication use | |
|---|---|
| Lithium Angiotensin II receptor blocker | |
| Anti-epileptic mood stabilizers | Angiotensin converting enzyme inhibitors |
| Anti-epileptics (other than mood stabilizers) | Beta blockers |
| Atypical antipsychotics | Calcium channel blockers |
| Benzodiazepines | Diuretics |
| Serotonin-norepinephrine reuptake Inhibitors | Nitrates |
| Selective serotonin reuptake inhibitors | Lipid lowering drugs |
| Tricyclic antidepressants (TCAs) | Non-insulin diabetes medications |
| Typical antipsychotics | Insulin |
| Anticoagulants | Antidepressants |
| Antiplatelet agents | |

| Rheumatoid arthritis related factors | |
|---|---|
| Number of combined biologic DMARDs (other than Use of other nonbiologic DMARDs) | |
| study medications) | |
| Number of combined nonbiologic DMARDs | Nonsteroidal anti-inflammatory drugs/COXIBs |
| Methotrexate | Glucocorticoid dose |
| Hydroxychloroquine | Opioids |
| Leflunomide | |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation Renal dysfunction | |
| Coronary artery disease | Chronic liver disease |
| Heart failure | Asthma |
| Stroke or transient ischemic attack | Ischemic heart disease |
| Peripheral vascular disease | Chronic obstructive pulmonary disease |

| Hypertension | Malignancy |
|----------------|-------------------------------------|
| Diabetes | Drug or alcohol abuse or dependence |
| Hyperlipidemia | Venous thromboembolism |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- **Primary outcome**: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:
   Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of tofacitinib and abatacept and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- · End of the study period,
- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (tofacitinib and abatacept) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of tofacitinib and abatacept and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

## 7. Feasibility counts

| Analysis scheme | Total<br>tofacitinib/abatacept<br>initiators | N outcome | Dementia Rate per 1,000<br>person-years (95% CI) | Follow-up time in days;<br>Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 4,456 (15.1%) | 316 | 7.05 (6.00, 0.71) | 224 [05, 500] |
| | 25,008 (84.9%) | 310 | 7.85 (6.98, 8.71) | 231 [86, 609] |
| 2: 6 mo induction period, 'as started' | 2,302 (12.9%) | F27 | 12.02 (12.74.15.00) | 1.044 [462, 1.005] |
| | 15,563 (87.1%) | 537 | 13.92 (12.74, 15.09) | 1,044 [463, 1,095] |
| 3: exclude 6 mo follow-up (symptoms to | 2,228 (12.6%) | 250 | 0.06 /7.01.10.10\ | 250 [121 910] |
| claims period) | 15,393 (87.1%) | 258 | 8.96 (7.91, 10.10) | 350 [121, 819] |
| 4: Outcome Dx + Rx | 4,456 (15.1%) | 122 | 2 20 (2 72 2 04) | 224 [05 544] |
| | 25,008 (84.9%) | 133 | 3.28 (2.73, 3.84) | 231 [86, 611] |

### 8. Propensity score analysis

We will use a propensity-score (PS)<sub>1</sub>-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.<sup>2</sup> Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,<sup>3</sup> and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.<sup>4</sup>

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups. Next, balance in each individual covariate between two treatment groups is reported using standardized differences.

# a. PS distributions stratified by treatment group

# Pre-matching propensity score overlap:



# Post-matching propensity score overlap:



# b. Table for covariate balance

| | | Unmatched | | | PS-Matched | |
|---|---|---|---|---|---|---|
| Variable | Tofacitinib<br>(N = 4,456) | Abatacept<br>(N = 25,008) | St. Diff | Tofacitinib<br>(N = 4,224) | Abatacept<br>(N = 4,224) | St. Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 72.11 (5.69) | 72.55 (5.81) | -0.08 | 72.18 (5.70) | 72.19 (5.59) | 0.00 |
| Gender, n (%) | | | | | | |
| Male | 778 (17.5%) | 4,426 (17.7%) | -0.01 | 751 (17.8%) | 752 (17.8%) | 0.00 |
| Female | 3,678 (82.5%) | 20,582 (82.3%) | 0.01 | 3,473 (82.2%) | 3,472 (82.2%) | 0.00 |
| Race, n (%) | | | | | | |
| White | 3,572 (80.2%) | 21,940 (87.7%) | -0.21 | 3,408 (80.7%) | 3,401 (80.5%) | 0.01 |
| Black | 488 (11.0%) | 1,506 (6.0%) | 0.18 | 442 (10.5%) | 434 (10.3%) | 0.01 |
| Asian | 96 (2.2%) | 311 (1.2%) | 0.08 | 92 (2.2%) | 97 (2.3%) | -0.01 |
| Hispanic | 138 (3.1%) | 675 (2.7%) | 0.02 | 132 (3.1%) | 137 (3.2%) | -0.01 |
| Native American | 30 (0.7%) | 116 (0.5%) | 0.03 | 27 (0.6%) | 28 (0.7%) | -0.01 |
| Other | 89 (2.0%) | 326 (1.3%) | 0.05 | 82 (1.9%) | 90 (2.1%) | -0.01 |
| Unknown | 43 (1.0%) | 134 (0.5%) | 0.06 | 41 (1.0%) | 37 (0.9%) | 0.01 |
| Region, n (%) | | | | | | |
| Northeast | 1,029 (23.1%) | 3,665 (14.7%) | 0.22 | 951 (22.5%) | 944 (22.3%) | 0.00 |
| South | 1,834 (41.2%) | 11,410 (45.6%) | -0.09 | 1,754 (41.5%) | 1,775 (42.0%) | -0.01 |
| North Central | 720 (16.2%) | 5,277 (21.1%) | -0.13 | 692 (16.4%) | 657 (15.6%) | 0.02 |
| West | 869 (19.5%) | 4,598 (18.4%) | 0.03 | 823 (19.5%) | 843 (20.0%) | -0.01 |
| Unknown | 4 (0.1%) | 58 (0.2%) | -0.03 | 4 (0.1%) | 5 (0.1%) | 0.00 |
| Calendar year of index date, n (%) | | | | | | |
| 2007 | 0 (0.0%) | 2,057 (8.2%) | -0.42 | 0 (0.0%) | 0 (0.0%) | 0.00 |
| 2008 | 0 (0.0%) | 1,814 (7.3%) | -0.40 | 0 (0.0%) | 0 (0.0%) | 0.00 |
| 2009 | 0 (0.0%) | 2,136 (8.5%) | -0.43 | 0 (0.0%) | 0 (0.0%) | 0.00 |

| 2010 | 0 (0.0%) | 1,959 (7.8%) | -0.41 | 0 (0.0%) | 0 (0.0%) | 0.00 |
|---|---|---|---|---|---|---|
| 2011 | 0 (0.0%) | 1,848 (7.4%) | -0.40 | 0 (0.0%) | 0 (0.0%) | 0.00 |
| 2012 | 15 (0.3%) | 2,249 (9.0%) | -0.42 | 15 (0.4%) | 17 (0.4%) | 0.00 |
| 2013 | 486 (10.9%) | 2,223 (8.9%) | 0.07 | 475 (11.2%) | 481 (11.4%) | -0.01 |
| 2014 | 850 (19.1%) | 2,133 (8.5%) | 0.31 | 807 (19.1%) | 831 (19.7%) | -0.02 |
| 2015 | 958 (21.5%) | 2,627 (10.5%) | 0.30 | 907 (21.5%) | 908 (21.5%) | 0.00 |
| 2016 | 903 (20.3%) | 2,808 (11.2%) | 0.25 | 859 (20.3%) | 840 (19.9%) | 0.01 |
| 2017 | 1,244 (27.9%) | 3,154 (12.6%) | 0.39 | 1,161 (27.5%) | 1,147 (27.2%) | 0.01 |
| Low income subsidy, n (%) | 1,600 (35.9%) | 4,409 (17.6%) | 0.42 | 1,396 (33.0%) | 1,383 (32.7%) | 0.01 |
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 1,411 (31.7%) | 7,583 (30.3%) | 0.03 | 1,338 (31.7%) | 1,329 (31.5%) | 0.00 |
| Obesity | 851 (19.1%) | 3,385 (13.5%) | 0.15 | 808 (19.1%) | 812 (19.2%) | 0.00 |
| Hypertension | 3,452 (77.5%) | 19,114 (76.4%) | 0.03 | 3,269 (77.4%) | 3,276 (77.6%) | 0.00 |
| Coronary artery disease | 1,166 (26.2%) | 6,837 (27.3%) | -0.02 | 1,111 (26.3%) | 1,138 (26.9%) | -0.01 |
| Depression | 933 (20.9%) | 4,678 (18.7%) | 0.06 | 876 (20.7%) | 855 (20.2%) | 0.01 |
| Anxiety | 769 (17.3%) | 3,243 (13.0%) | 0.12 | 717 (17.0%) | 706 (16.7%) | 0.01 |
| Bipolar disorder | 49 (1.1%) | 241 (1.0%) | 0.01 | 44 (1.0%) | 53 (1.3%) | -0.03 |
| Schizophrenia | 16 (0.4%) | 33 (0.1%) | 0.06 | 10 (0.2%) | 12 (0.3%) | -0.02 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 1,187 (26.6%) | 4,485 (17.9%) | 0.21 | 1,116 (26.4%) | 1,130 (26.8%) | -0.01 |
| Mammography, n (%) | 1,488 (33.4%) | 8,205 (32.8%) | 0.01 | 1,415 (33.5%) | 1,390 (32.9%) | 0.01 |
| Colonoscopy, n (%) | 452 (10.1%) | 3,146 (12.6%) | -0.08 | 434 (10.3%) | 412 (9.8%) | 0.02 |
| Fecal occult blood test, n (%) | 383 (8.6%) | 2,401 (9.6%) | -0.03 | 367 (8.7%) | 369 (8.7%) | 0.00 |
| Influenza vaccination, n (%) | 2,928 (65.7%) | 17,111 (68.4%) | -0.06 | 2,791 (66.1%) | 2,772 (65.6%) | 0.01 |
| Pneumococcal vaccination, n (%) | 1,819 (40.8%) | 6,599 (26.4%) | 0.31 | 1,717 (40.6%) | 1,701 (40.3%) | 0.01 |
| Herpes zoster vaccination, n (%) | 32 (0.7%) | 122 (0.5%) | 0.03 | 25 (0.6%) | 26 (0.6%) | 0.00 |
| Bone mineral density test, n (%) | 1,103 (24.8%) | 7,761 (31.0%) | -0.14 | 1,060 (25.1%) | 1,092 (25.9%) | -0.02 |

| Number of distinct generic agents, mean (SD) | 15.99 (7.23) | 14.51 (6.69) | 0.00 | 15.81 (7.11) | 15.95 (7.40) | 0.00 |
|---|---|---|---|---|---|---|
| Number of emergency room visits, mean (SD) | 0.69 (1.38) | 0.65 (1.18) | 0.00 | 0.69 (1.37) | 0.70 (1.28) | 0.00 |
| Number of outpatient visits, mean (SD) | 18.73 (19.02) | 20.75 (17.93) | 0.00 | 18.77 (19.30) | 18.95 (14.06) | 0.00 |
| Number of hospitalizations, mean (SD) | 0.31 (0.84) | 0.36 (0.79) | 0.00 | 0.31 (0.84) | 0.31 (0.73) | 0.00 |
| Number of physician office visits, mean (SD) | 4.92 (9.57) | 5.53 (8.58) | 0.00 | 4.92 (9.75) | 5.00 (6.31) | 0.00 |
| Number of rheumatologist visits, mean (SD) | 4.39 (3.15) | 5.44 (4.06) | 0.00 | 4.44 (3.16) | 4.49 (3.14) | 0.00 |
| Number of C-reactive protein tests ordered, mean (SD) | 2.56 (2.29) | 2.79 (2.70) | 0.00 | 2.59 (2.30) | 2.61 (2.34) | 0.00 |
| Number of serum creatinine tests ordered, mean (SD) | 5.81 (3.38) | 6.59 (3.62) | 0.00 | 5.87 (3.42) | 5.95 (3.18) | 0.00 |
| Composite frailty score, mean (SD) | 0.17 (0.04) | 0.17 (0.04) | 0.00 | 0.17 (0.04) | 0.17 (0.04) | 0.00 |
| Osteoporosis, n (%) | 1,734 (38.9%) | 10,744 (43.0%) | -0.08 | 1,637 (38.8%) | 1,669 (39.5%) | -0.01 |
| Fractures, n (%) | 499 (11.2%) | 2,762 (11.0%) | 0.01 | 465 (11.0%) | 499 (11.8%) | -0.03 |
| Falls, n (%) | 215 (4.8%) | 1,188 (4.8%) | 0.00 | 207 (4.9%) | 205 (4.9%) | 0.00 |
| Use of supplemental oxygen, n (%) | 101 (2.3%) | 322 (1.3%) | 0.08 | 90 (2.1%) | 77 (1.8%) | 0.02 |
| Combined comorbidity score, mean (SD) | 1.59 (2.24) | 1.58 (2.23) | 0.00 | 1.60 (2.26) | 1.61 (2.25) | 0.00 |
| Comedication use, n (%) | | | | | | |
| Lithium | 9 (0.2%) | 24 (0.1%) | 0.03 | 6 (0.1%) | 6 (0.1%) | 0.00 |
| Anti-epileptic mood stabilizers | 68 (1.5%) | 315 (1.3%) | 0.02 | 64 (1.5%) | 73 (1.7%) | -0.02 |
| Anti-epileptics (other than mood stabilizers) | 1,261 (28.3%) | 6,063 (24.2%) | 0.09 | 1,187 (28.1%) | 1,192 (28.2%) | 0.00 |
| Atypical antipsychotics | 110 (2.5%) | 368 (1.5%) | 0.07 | 93 (2.2%) | 93 (2.2%) | 0.00 |
| Benzodiazepines | 978 (21.9%) | 3,068 (12.3%) | 0.26 | 920 (21.8%) | 935 (22.1%) | -0.01 |
| Serotonin-norepinephrine reuptake inhibitors | 626 (14.0%) | 2,818 (11.3%) | 0.08 | 583 (13.8%) | 581 (13.8%) | 0.00 |

| Selective serotonin reuptake inhibitors | 879 (19.7%) | 5,133 (20.5%) | -0.02 | 835 (19.8%) | 818 (19.4%) | 0.01 |
|---|---|---|---|---|---|---|
| Tricyclic antidepressants (TCAs) | 268 (6.0%) | 1,883 (7.5%) | -0.06 | 252 (6.0%) | 256 (6.1%) | 0.00 |
| Typical antipsychotics | 7 (0.2%) | 52 (0.2%) | 0.00 | 6 (0.1%) | 4 (0.1%) | 0.00 |
| Anticoagulants | 472 (10.6%) | 2,718 (10.9%) | -0.01 | 449 (10.6%) | 455 (10.8%) | -0.01 |
| Antiplatelet agents | 367 (8.2%) | 2,204 (8.8%) | -0.02 | 346 (8.2%) | 351 (8.3%) | 0.00 |
| Angiotensin II receptor blockers | 1,137 (25.5%) | 5,856 (23.4%) | 0.05 | 1,079 (25.5%) | 1,078 (25.5%) | 0.00 |
| Angiotensin converting enzyme inhibitors | 1,182 (26.5%) | 7,120 (28.5%) | -0.04 | 1,115 (26.4%) | 1,133 (26.8%) | -0.01 |
| Beta blockers | 1,777 (39.9%) | 9,906 (39.6%) | 0.01 | 1,690 (40.0%) | 1,717 (40.6%) | -0.01 |
| Calcium channel blockers | 1,313 (29.5%) | 6,972 (27.9%) | 0.04 | 1,242 (29.4%) | 1,213 (28.7%) | 0.02 |
| Diuretics | 1,397 (31.4%) | 8,277 (33.1%) | -0.04 | 1,329 (31.5%) | 1,329 (31.5%) | 0.00 |
| Nitrates | 298 (6.7%) | 1,775 (7.1%) | -0.02 | 283 (6.7%) | 294 (7.0%) | -0.01 |
| Lipid lowering drugs | 2,245 (50.4%) | 11,919 (47.7%) | 0.05 | 2,125 (50.3%) | 2,191 (51.9%) | -0.03 |
| Non-insulin diabetes medications | 752 (16.9%) | 3,880 (15.5%) | 0.04 | 710 (16.8%) | 682 (16.1%) | 0.02 |
| Insulin | 307 (6.9%) | 1,484 (5.9%) | 0.04 | 290 (6.9%) | 290 (6.9%) | 0.00 |
| Antidepressants | 1,776 (39.9%) | 9,580 (38.3%) | 0.03 | 1,677 (39.7%) | 1,665 (39.4%) | 0.01 |
| Rheumatoid arthritis related factors | | | | | | |
| Number of combined biologic<br>DMARDs, n (%) | | | | | | |
| 0 | 1,532 (34.4%) | 8,780 (35.1%) | -0.01 | 1,454 (34.4%) | 1,417 (33.5%) | 0.02 |
| 1 | 1,578 (35.4%) | 11,711 (46.8%) | -0.23 | 1,513 (35.8%) | 1,514 (35.8%) | 0.00 |
| 2 | 922 (20.7%) | 3,566 (14.3%) | 0.17 | 866 (20.5%) | 873 (20.7%) | 0.00 |
| 3 or more | 424 (9.5%) | 951 (3.8%) | 0.23 | 391 (9.3%) | 420 (9.9%) | -0.02 |
| Number of combined nonbiologic DMARDs, n (%) | | | | | | |
| 0 | 420 (9.4%) | 2,363 (9.4%) | 0.00 | 396 (9.4%) | 416 (9.8%) | -0.01 |
| 1 | 1,613 (36.2%) | 10,332 (41.3%) | -0.10 | 1,542 (36.5%) | 1,494 (35.4%) | 0.02 |
| 2 | 1,398 (31.4%) | 7,573 (30.3%) | 0.02 | 1,312 (31.1%) | 1,311 (31.0%) | 0.00 |

| 3 or more | 1,025 (23.0%) | 4,740 (19.0%) | 0.10 | 974 (23.1%) | 1,003 (23.7%) | -0.01 |
|---|---|---|---|---|---|---|
| Use of other nonbiologic DMARDs, n (%) | 868 (19.5%) | 4,432 (17.7%) | 0.05 | 817 (19.3%) | 875 (20.7%) | -0.04 |
| Methotrexate, n (%) | 2,279 (51.1%) | 14,395 (57.6%) | -0.13 | 2,168 (51.3%) | 2,129 (50.4%) | 0.02 |
| Hydroxychloroquine, n (%) | 1,095 (24.6%) | 5,885 (23.5%) | 0.03 | 1,038 (24.6%) | 1,070 (25.3%) | -0.02 |
| Leflunomide, n (%) | 953 (21.4%) | 4,742 (19.0%) | 0.06 | 902 (21.4%) | 888 (21.0%) | 0.01 |
| Nonsteroidal anti-inflammatory drugs/Coxibs, n (%) | 1,578 (35.4%) | 8,423 (33.7%) | 0.04 | 1,474 (34.9%) | 1,472 (34.8%) | 0.00 |
| Opioids, n (%) | 3,033 (68.1%) | 18,062 (72.2%) | -0.09 | 2,870 (67.9%) | 2,877 (68.1%) | 0.00 |
| Glucocorticoids use/dose, n (%) | 3,292 (73.9%) | 18,512 (74.0%) | 0.00 | 3,127 (74.0%) | 3,099 (73.4%) | 0.01 |
| Comorbid conditions, n (%) | | | | | | |
| Atrial fibrillation | 464 (10.4%) | 2,908 (11.6%) | -0.04 | 451 (10.7%) | 435 (10.3%) | 0.01 |
| Heart failure | 543 (12.2%) | 3,212 (12.8%) | -0.02 | 522 (12.4%) | 526 (12.5%) | 0.00 |
| Stroke or transient ischemic attack | 360 (8.1%) | 2,233 (8.9%) | -0.03 | 343 (8.1%) | 343 (8.1%) | 0.00 |
| Peripheral vascular disease | 570 (12.8%) | 3,051 (12.2%) | 0.02 | 542 (12.8%) | 537 (12.7%) | 0.00 |
| Hyperlipidemia | 2,978 (66.8%) | 16,683 (66.7%) | 0.00 | 2,824 (66.9%) | 2,834 (67.1%) | 0.00 |
| Renal dysfunction | 748 (16.8%) | 3,774 (15.1%) | 0.05 | 721 (17.1%) | 723 (17.1%) | 0.00 |
| Chronic liver disease | 374 (8.4%) | 2,402 (9.6%) | -0.04 | 361 (8.5%) | 362 (8.6%) | 0.00 |
| Asthma | 1,003 (22.5%) | 4,028 (16.1%) | 0.16 | 940 (22.3%) | 939 (22.2%) | 0.00 |
| Ischemic heart disease | 1,135 (25.5%) | 6,650 (26.6%) | -0.03 | 1,080 (25.6%) | 1,103 (26.1%) | -0.01 |
| Chronic obstructive pulmonary disease | 1,213 (27.2%) | 6,165 (24.7%) | 0.06 | 1,135 (26.9%) | 1,111 (26.3%) | 0.01 |
| Malignancy | 926 (20.8%) | 6,219 (24.9%) | -0.10 | 901 (21.3%) | 904 (21.4%) | 0.00 |
| Drug or alcohol abuse or dependence | 535 (12.0%) | 1,795 (7.2%) | 0.16 | 490 (11.6%) | 480 (11.4%) | 0.01 |
| Venous thromboembolism | 261 (5.9%) | 1,453 (5.8%) | 0.00 | 243 (5.8%) | 249 (5.9%) | 0.00 |

### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

### 10. References

- 1. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 5. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. Comp Effect Res 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- 7. Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.

| # | Implementation in routine care | |
|---|---|---|
| | | EXPOSURE vs. COMPARISON |
| | Tofacitinib vs Abatacept | |
| | | INCLUSION CRITERIA |
| 1 | No prior use of tofacitinib or abatacept | Depending on the comparison group, we will require new-use (defined as no use anytime prior to index date) of tofacitinib and abatacept |
| 2 | Sufficient enrollment | Medicare Part A, B, and D enrollment with no HMO coverage for 365 days prior to and on the cohort entry date |
| | | EXCLUSION CRITERIA |
| | Prior history of dementia | Measured any time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| | | ICD9 diagnosis – 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 ICD10 diagnosis – F01.xx-F03.xx, G30.xx-G31.85, R41.xx |
| 1 | | NDC brand name – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or "REMINYL" |
| | | NDC generic name – "DONEPEZIL HCL", "GALANTAMINE HBR", "MEMANTINE HCL", "MEMANTINE HCL/DONEPEZIL HCL", "RIVASTIGMINE", or "RIVASTIGMINE TARTRATE" |
| | No prior history of rheumatoid arthritis | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| 2 | | ICD9 diagnosis – 714.xx<br>ICD10 diagnosis – M05.xx, M06.xx, M08.xx, M12.xx |
| | Nursing home admission | Measured 365 days prior to drug initiation – |
| 3 | | MEDPAR - Short Stay/Long Stay/SNF Indicator Code – N = SNF Stay (Prvdr3 = 5, 6, U, W, Y, or Z) |

| Covariate list | |
|---|---|
| | Potential confounders |
| Category | ICD-9 |
| | Age |
| | Gender |
| | Race |
| Demographics | Region |
| | Calendar year of index date |
| | Low income subsidy |
| | , |
| | Diabetes |
| | Obesity |
| | Hypertension |
| | Coronary artery disease |
| Dementia risk factors | Depression |
| | Anxiety |
| | Bipolar disorder |
| | Schizophrenia |
| | Sunzopin cinu |
| | Smoking |
| | Mammography |
| | Colonoscopy |
| | Fecal occult blood test |
| Lifestyle factors and markers for healthy behavior | Influenza vaccination |
| | Pneumococcal vaccination |
| | Herpes zoster vaccination |
| | BMD test |
| | BIVID LEST |
| | Number of distinct generic agents |
| | Number of distinct generic agents Number of emergency room visits |
| | Number of outpatient visits |
| | Number of outpatient visits Number of hospitalizations |
| Healthcare utilization measures | Number of physician office visits |
| | Number of rheumatologist visits Number of CRP tests ordered |
| | Number of CRP tests ordered Number of serum creatinine tests ordered |
| | Number of serum creatifine tests ordered |
| | Company C. III |
| | Composite frailty score |
| | Osteoporosis |
| Frailty markers | Fractures |
| | Falls |
| | Use of supplemental oxygen |
| | A combined comorbidity score |
| RA-specific como | |
| | Lithium |
| | Anti-epileptic mood stabilizers |
| | Anti-epileptics (other than mood stabilizers) |

| | Atypical antipsychotics |
|---|---|
| | Benzodiazepines |
| | SNRIs |
| | SSRIs |
| | TCAs |
| | Typical antipsychotics |
| | Anticoagulants |
| Comedications | Antiplatelet agents |
| | Angiotensin II receptor blockers |
| | Angiotensin converting enzyme inhibitors |
| | Beta blockers |
| | Calcium channel blockers |
| | Diuretics |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | инисрессовно |
| | Number of biologic DMARDs |
| | Number of nonbiologic DMARDs |
| | Use of other nonbiologic DMARDs |
| | Methotrexate |
| | Hydroxychloroguine |
| | Leflunomide |
| | Sulfasalazine |
| Nonbiologics | Anakinra |
| | Auranofin |
| | Azathioprine |
| | Cyclosporine |
| | Cyclosphosphamide |
| | Gold sodium thiomalate |
| | NSAID/COXIB |
| | Opioids |
| | Glucocorticoids |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Hypertension |
| | Diabetes |
| | Hyperlipidemia |
| Com orbid conditions | |
| Com orbid conditions | Hyperlipidemia Renal dysfunction Chronic liver disease |
| Com orbid conditions | Renal dysfunction |

# Appendix A

| • | |
|---|-------------------------------------|
| | COPD |
| | Malignancy |
| | Drug or alcohol abuse or dependence |
| | VTE |

# Appendix A Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2007 |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |

### Low income subsidy

https://www.cms.gov/Medicare/Eligibility-and-

 $\underline{Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pdf}$ 

#### Diabetes


#### Obesity


### Prescriptions

Orlistat
Sibutramine
Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

Hypertension

| Hypertension | | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
| I10 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| I10 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| I160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| l161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| I110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| I110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, malignant, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | kidney disease stage I through stage IV, or unspecified |
| | | disease | |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | stage renal disease | or end stage renal disease |

| I1310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
|---|---|---|---|
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| 1150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| l151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| l152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| 1158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| 1159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

Coronary artery disease


| eral wall, initial<br>eral wall, subsequent<br>sterior wall, episode |
|----------------------------------------------------------------------|
| sterior wall, episode |
| sterior wall, initial |
| sterior wall, initial |
| sterior wall, |
| ferior wall, episode of |
| ferior wall, initial |
| ferior wall, initial |
| ferior wall, |
| teral wall, episode of |
| teral wall, initial |
| teral wall, initial |
| teral wall, |
| of care unspecified |
| pisode of care |
| oisode of care |
| ent episode of care |
| are unspecified |
| • |
| de of care |
| de of care |
| episode of care |
| ecified sites, episode |
| ecified sites, initial |
| , |
| ecified sites, initial |
| ecified sites, initial |
| ecified sites, |
| ied site, episode of |
| ied site, initial |
| ied site, initial |
| ied site, subsequent |
| tuno of |
| type of vessel, |


Depression


#### Anxiety


#### Bipolar disorder


# Appendix A Dementia risk factors


#### Schizophrenia


### Smoking


OR dispensing of: At least one nicotine or varenicline prescription

## Mammography


Colonoscopy


49

Appendix A Lifestyle factors and markers for healthy behavior

| 45380 |
|-------|
| 45381 |
| 45382 |
| 45383 |
| 45384 |
| 45385 |
| 45386 |
| 45387 |
| 45388 |
| 45389 |
| 45390 |
| 45391 |
| 45392 |
| HCPCS |
| G0105 |
| G0121 |

### Fecal occult blood test


### Influenza vaccination


#### Pneumococcal vaccination


50

Appendix A Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

### Herpes zoster vaccination


#### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

#### Healthcare utilization measures

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

#### Number of rheumatologist visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

66 = Rheumatology (eff 5/92) Note: during 93/94 DMERC also used this to mean medical supply company with respiratory therapist

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99000 | 99141 | 99249 | 99347 | 99450 | 99603 |
| 99001 | 99142 | 99250 | 99348 | 99454 | 99604 |
| 99002 | 99143 | 99251 | 99349 | 99455 | 99605 |
| 99003 | 99144 | 99252 | 9934S | 99456 | 99606 |
| 99004 | 99145 | 99253 | 99350 | 99460 | 99607 |
| 99005 | 99148 | 99254 | 99351 | 99461 | 99615 |
| 99006 | 99149 | 99255 | 99352 | 99462 | 99649 |
| 99010 | 09915 | 99256 | 99353 | 99463 | 99675 |
| 99011 | 99150 | 9925S | 99354 | 99464 | 99684 |
| 99012 | 99160 | 99261 | 99355 | 99465 | 99700 |
| 99014 | 99163 | 99262 | 99356 | 99466 | 99703 |
| 99015 | 99166 | 99263 | 99357 | 99467 | 99707 |
| 99020 | 99170 | 99270 | 99358 | 99468 | 99713 |
| 99023 | 99171 | 99271 | 99359 | 99469 | 99714 |

| 99024 99172 99272 99350 99471 99737 99025 99173 99274 99360 99471 99732 99026 99174 99274 99361 99475 99762 99027 99175 99275 99362 99475 99762 99028 99178 99280 99363 99476 99770 99032 99183 99280 99363 99477 99770 99032 99183 99281 99364 99477 99772 99038 99184 99282 99365 99478 99776 99038 99185 99284 99367 99479 99780 99039 99186 99284 99367 99480 99799 99040 99188 99284 99367 99480 99799 99041 99180 99286 99371 99482 99381 99041 99190 99286 99371 99485 99801 99042 99191 99288 99373 99485 99802 99047 99195 99288 99373 99486 99803 99048 99199 99200 99375 99487 99806 99049 99049 99191 99289 99376 99489 99810 99049 99049 99200 99375 99489 99810 99051 99200 99292 99377 99489 99810 99051 99200 99292 99377 99489 99811 99051 99200 99292 99377 99489 99811 99052 99203 99378 99495 99383 99384 99810 99054 99200 99292 99377 99489 99811 99059 99009 99200 99399 99399 99399 99381 99309 99009 99200 99399 993999 99399 993999 99399 9939 | | | | | | |
|---|---|---|---|---|---|---|
| 99026 99174 99274 99361 99475 9976 99776 99027 99178 99280 99362 99475 99770 99028 99178 99280 99383 99476 99770 99032 99183 99281 99384 99282 99385 99478 99776 99038 99188 99282 99385 99478 99776 99038 99188 99282 99385 99478 99776 99038 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99799 99040 99180 99180 99286 99371 99482 99801 99062 99180 99286 99371 99482 99801 99062 99180 99286 99371 99485 99801 99062 99192 99288 99284 99377 99485 99802 99063 99244 99390 99388 99377 99485 99802 99064 99192 99289 99274 99485 99803 99284 99379 99485 99803 99284 99379 99485 99803 99280 99377 99485 99803 99280 99378 99388 99377 99485 99802 99378 99388 99389 99388 99389 99388 99389 99388 99389 99388 99389 99388 99389 99388 99389 99389 99388 99389 99388 99389 99388 99389 9 | 99024 | 99172 | 99272 | 9935D | 99470 | 99717 |
| 99027 99175 99275 99362 99475 99762 997028 99178 992028 99178 99203 99318 99281 99365 99476 99777 99772 99035 99183 99281 99365 99476 99776 99772 99035 99184 99283 99366 99479 99780 99036 99185 99283 99366 99479 99780 99039 99185 99283 99366 99479 99780 99039 99186 99284 99367 99480 99799 99780 99040 99188 99286 99285 99366 99479 99780 99040 99188 99286 99287 99372 99486 99801 99286 99371 99482 99801 99286 99371 99482 99801 99286 99373 99486 99803 99047 99195 99289 99373 99486 99803 99047 99195 99290 99375 99488 99810 99049 99200 99291 99376 99488 99811 99060 99291 99376 99488 99811 99060 99291 99376 99489 99814 99051 99202 99293 99378 99496 99831 99060 99201 99202 99377 99490 99381 99060 99201 99202 99378 99496 99831 99060 99206 99206 99206 99206 99206 99206 99380 99349 99360 99360 99206 99206 99206 99380 99349 99380 99349 99360 99360 99206 9920 | 99025 | 99173 | 99273 | 99360 | 99471 | 99732 |
| 99027 99175 99275 99362 99475 99762 997028 99178 992028 99178 99203 99318 99281 99365 99476 99777 99772 99035 99183 99281 99365 99476 99776 99772 99035 99184 99283 99366 99479 99780 99036 99185 99283 99366 99479 99780 99039 99185 99283 99366 99479 99780 99039 99186 99284 99367 99480 99799 99780 99040 99188 99286 99285 99366 99479 99780 99040 99188 99286 99287 99372 99486 99801 99286 99371 99482 99801 99286 99371 99482 99801 99286 99373 99486 99803 99047 99195 99289 99373 99486 99803 99047 99195 99290 99375 99488 99810 99049 99200 99291 99376 99488 99811 99060 99291 99376 99488 99811 99060 99291 99376 99489 99814 99051 99202 99293 99378 99496 99831 99060 99201 99202 99377 99490 99381 99060 99201 99202 99378 99496 99831 99060 99206 99206 99206 99206 99206 99206 99380 99349 99360 99360 99206 99206 99206 99380 99349 99380 99349 99360 99360 99206 9920 | 99026 | 99174 | 99274 | 99361 | 99472 | 99736 |
| 99028 99178 99280 99364 99477 99770 99032 99184 99281 99364 99477 99770 99035 99184 99282 99365 99478 99776 99038 99186 99282 99365 99478 99776 99038 99186 99284 93667 99480 99776 99038 99186 99284 93667 99480 99779 99041 99180 99286 99371 99482 99780 99041 99191 99287 99286 99371 99482 993602 99045 99191 99287 99288 99373 99485 99302 99045 99195 99289 99373 99485 99302 99045 99195 99289 99374 99487 99806 99049 99049 99195 99290 99375 99488 99374 99488 99311 99049 99200 9921 99376 99488 99373 99496 99200 99201 99376 99488 99381 99059 99202 99203 99377 99490 99381 99381 99059 99202 99203 99377 99490 99381 99381 99059 99202 99203 99379 99496 99381 99059 99206 99206 99206 99209 99379 99496 99389 | | | | | | |
| 99032 99183 99281 99364 99477 99772 99035 99184 99282 99365 99478 99776 99038 99185 99284 99367 99480 99780 99039 99186 99284 99367 99480 99799 99039 99186 99285 99368 99481 9979A 99041 99190 99286 99271 99482 99381 99041 99190 99286 99271 99482 99382 99042 99111 99286 99271 99485 99801 99043 99191 99286 99271 99485 99802 99047 99195 99288 99374 99485 99803 99047 99195 99288 99374 99487 99803 99049 99190 99290 99375 99488 99810 99049 99200 99291 99376 99489 99811 99050 99201 99292 99377 99490 99381 99051 99202 99293 99378 99496 99383 99054 99205 99296 99381 99494 99399 99054 99206 99296 99381 99498 99841 99056 99206 99296 99381 99498 99841 99056 99207 99298 99382 99499 99884 99058 99207 99298 99383 99500 99894 99060 99208 9930 99385 99500 99894 99060 99208 9930 99385 99500 99894 99060 99208 9930 99385 99500 99894 99070 99208 9930 99385 99502 99899 99060 99208 9930 99385 99502 99899 99071 99208 9930 99387 99506 99899 99071 99208 9930 99387 99506 99899 99071 99208 9930 99387 99506 99899 99071 99208 9930 99387 99506 99899 99071 99208 9930 99384 99501 99897 99072 99210 9930 99385 99502 99899 99073 99208 9930 99385 99502 99899 99074 99210 99303 99397 99505 99301 99307 99075 99210 99303 99307 99307 99307 99307 99307 99307 99308 99309 | | | | | | |
| 99035 99184 99282 99365 99478 99776 99038 99186 99284 99366 9477 99780 99039 99186 99284 99367 99480 99799 99030 99186 99284 99367 99480 99799 99040 99188 99285 99368 9481 99793 99041 99190 99286 9271 99482 99801 99042 99191 99287 99372 39485 99802 99043 99195 99288 99373 99486 99802 99044 99195 99289 99374 99487 99806 99048 99199 99290 99375 99488 99811 99049 99200 99201 99376 99488 99811 99050 99201 99376 99489 99811 99050 99201 99377 99490 99381 99051 99202 9923 99377 99490 99814 99051 99202 9923 99377 99490 99814 99052 99204 99295 99380 99495 99821 99053 99204 99295 99380 99497 99880 99881 99054 99206 99296 99381 99498 99841 99056 99206 99297 99382 99499 99881 99840 99058 99206 99297 99382 99499 99881 99841 99058 99206 99297 99382 99499 99881 99806 99060 99201 99200 99201 99379 99496 99881 99058 99206 99207 99382 99379 99498 99841 99058 99206 99207 99382 99498 99841 99058 99206 99207 99382 99499 99881 99058 99207 99382 99389 | | | | | | |
| 99038 99186 99284 99367 99480 99799 9040 99188 99285 92368 99480 99799 9041 99180 99286 92371 99482 99301 9042 99191 99286 99371 99482 99801 9042 99191 99288 99373 99485 99803 9044 99192 99288 99373 99486 99803 9047 99195 99288 99374 99487 99803 9048 99199 99290 99375 99488 99810 9008 99199 99290 99375 99488 99810 9008 99199 99290 99375 99488 99810 9008 99201 99292 99377 99480 99814 9009 99201 99292 99377 99480 99814 9001 99202 99293 99378 99495 99821 9002 99203 99294 99377 99490 99814 9005 99206 99206 99380 99497 99848 9008 99199 99206 99389 99496 99881 9009 99200 99209 99378 99496 99883 9001 99200 99209 99378 99496 99881 99811 9002 99208 99206 99389 99497 99849 99841 9005 99206 99206 99389 99389 99497 99881 9006 99207 99208 99389 99389 99499 99881 9006 99208 99209 99389 99389 99499 99881 9006 99208 99209 99309 99389 99499 99881 9006 99208 99209 99309 99384 99500 99894 9006 99208 99209 99309 99384 99500 99884 9006 99208 99209 99309 99384 99500 99884 9006 99208 99209 99309 99384 99500 99884 9007 99208 99309 99385 99500 99809 9007 99208 99309 99385 99500 99809 9007 99208 99300 99386 99503 99501 9007 99208 99300 99386 99503 99501 9007 99208 99300 99386 99503 99501 9007 99208 99309 99309 99309 99500 99007 90071 09921 99302 99301 99302 99309 9007 99208 99309 99309 99309 99500 99007 90072 99210 99302 99309 99309 99500 99007 90073 99211 99304 99309 99309 99500 99010 90074 99211 99304 99309 99309 99500 99010 90075 99212 99306 99309 99309 99500 99010 90079 99213 99306 99309 99309 99500 99010 90079 99215 99309 99308 99309 99500 99910 90079 99215 99309 99308 99309 99500 99910 90079 99215 99309 99308 99309 99500 99910 90079 99215 99309 99308 99309 99500 99910 90079 99215 99309 99309 99309 99500 99900 99000 99000 99216 99300 993 | | | | | | |
| 99033 99186 99285 99386 99481 99799 99001 99188 99285 99386 99481 99799 99001 99188 99286 99371 99482 99801 99042 99191 99286 99371 99485 99803 99043 99191 99288 99373 99485 99806 99047 99195 99288 99373 99486 99803 99047 99195 99288 99373 99486 99806 99048 99199 99290 99376 99488 99377 99488 99381 99048 99199 99200 99291 99376 99489 99811 99050 99200 99291 99376 99489 99811 99050 99202 99293 99378 99495 99495 99495 99495 99496 99505 99204 99292 99378 99496 99497 99406 99295 99296 99383 99497 99406 99295 99296 99383 99497 99406 99295 99296 99383 99497 99406 99296 99296 99383 99498 99498 99406 99296 99299 99383 99500 99296 99385 99206 99296 99383 99500 99296 99385 99500 99296 99385 99500 99296 99296 99385 99500 99596 99296 99385 99500 99596 99386 99500 99200 99299 99383 99500 99596 99386 99500 99296 99386 99500 99596 99386 99500 99596 | 99035 | 99184 | 99282 | 99365 | 99478 | 99776 |
| 99040 99188 99285 99388 99481 9979A 99001 99041 99191 99286 99771 99485 99802 99191 99287 99288 99273 99486 99802 99047 99191 99288 99273 99486 99802 99047 99195 99288 99274 99487 99806 99806 99003 99047 99195 99289 99374 99487 99886 99806 99008 99009 99290 99290 99375 99488 99810 99009 99009 99290 99290 99376 99489 99811 99000 99291 99376 99489 99811 99000 99291 99376 99490 99814 99000 99291 99377 99490 99814 99000 99290 99290 99378 99496 99833 990052 99203 99294 99379 99389 99496 99833 99055 99206 99206 99206 99206 99206 99207 99295 99380 99497 99884 99006 99206 99206 99296 99381 99498 99498 99881 99056 99206 99206 99296 99381 99499 99881 99066 99208 99299 99384 99500 99894 99060 99208 99296 99386 99207 99296 99386 99207 99298 99399 99399 99390 99390 99390 9930 99207 99298 9930 9930 9930 9930 9930 9930 9930 99 | 99038 | 99185 | 99283 | 99366 | 99479 | 99780 |
| 99040 99188 99285 99388 99481 9979A 99001 99041 99191 99286 99771 99485 99802 99191 99287 99288 99273 99486 99802 99047 99191 99288 99273 99486 99802 99047 99195 99288 99274 99487 99806 99003 99047 99195 99289 99374 99487 99806 99008 99009 99290 99290 99290 99375 99488 99810 99009 99009 99290 99290 99376 99489 99811 990051 99200 99291 99376 99499 99811 990051 99200 99291 99377 99490 99814 990051 99200 99292 99377 99490 99814 990052 99203 99203 99294 99378 99496 99833 99052 99205 99206 99295 99380 99496 99833 99056 99206 99206 99295 99380 99497 99884 99056 99206 99206 99206 99296 99381 99498 99881 99056 99206 99206 99296 99381 99498 99881 99066 99208 99296 99381 99498 99881 99066 99208 99296 99381 99498 99881 99066 99208 99296 99386 99207 99298 99399 99399 99399 99399 99390 9930 99296 9930 9930 9930 9930 9930 9930 9930 99 | 99039 | 99186 | 99284 | 99367 | 99480 | 99799 |
| 99041 99190 99287 99371 99482 99801 99042 99191 99287 99372 99486 99803 99047 99192 99288 99373 99486 99803 99047 99195 99288 99374 99486 99803 99048 99199 99290 99375 99488 99810 99048 99199 99290 99375 99488 99810 99049 99000 99291 99376 99489 99811 99050 99200 99291 99376 99489 99811 99050 99200 99292 99377 99490 99381 99050 99202 99293 99378 99495 99821 99052 99293 99378 99495 99821 99052 99293 99378 99495 99821 99052 99293 99378 99496 99821 99056 99206 99293 99380 99497 99494 99381 99056 99206 99297 99382 99380 99497 99494 99381 99056 99206 99297 99383 99499 99881 99058 99206 99297 99383 99499 99881 99058 99206 99297 99383 99499 99881 99058 99206 99299 99380 99399 99300 | | | | | | |
| 99042 99191 99288 99372 99485 99802 99045 99192 99288 99374 99486 99802 99047 99195 99288 99374 99487 99806 99049 99199 99290 99375 99488 99811 99049 99200 99291 99375 99488 99811 99059 99291 99376 99489 99811 99051 99292 99377 99490 98814 99051 99202 99292 99377 99490 98814 99051 99203 99203 99293 99378 99496 99881 99052 99203 99204 99292 99378 99496 99833 99053 99204 99295 99380 99496 99833 99205 99205 99206 99295 99380 99497 99496 99831 99205 99206 99297 99380 99498 99498 99491 99056 99206 99206 99297 99382 99499 99881 99056 99206 99297 99383 99500 99206 99299 99384 99501 99897 99003 99208 99299 99384 99501 99897 99003 99208 99299 99384 99501 99897 99003 99208 99209 99390 99386 99500 99209 9930 9930 9930 9930 9930 9930 9 | | | | | | |
| 99045 99192 99288 99373 99486 99803 99047 99195 99299 99299 99375 99487 99806 99009 99299 99299 99375 99488 99810 99009 99200 99291 99376 99489 99811 99050 99376 99489 99811 99050 99202 99293 99378 99495 99812 99051 99062 99293 99378 99495 99812 99052 99293 99378 99495 99812 99052 99293 99378 99496 99814 99052 99293 99294 99379 99496 99833 99064 99295 99296 99381 99496 99833 99065 99206 99296 99381 99498 99414 99056 99206 99296 99383 99499 99506 99296 99383 99500 99894 99006 99297 99382 99383 99500 99894 99006 99299 9930 99385 99500 99899 9930 9930 9930 99385 99502 99899 9930 9930 9930 99385 99502 99899 99006 99200 99300 99385 99502 99899 99007 99200 99300 99385 99502 99899 99007 99200 99300 99385 99502 99899 99007 99200 99300 99385 99506 99506 99007 99200 99300 99385 99506 99506 99007 99007 99200 99300 99300 99385 99506 99907 99007 99200 99300 99300 99385 99500 99910 99007 99200 99300 99300 99385 99500 99910 99007 99200 99300 99300 99386 99500 99910 99007 99200 99300 99300 99386 99500 99910 99007 99200 99300 99300 99386 99500 99910 99007 99200 99300 99300 99338 99500 99910 99007 99210 99303 99303 99300 99338 99506 99910 99007 99210 99303 99303 99506 99911 99007 99210 99303 99303 99506 99911 99007 99210 99303 99305 99506 99911 99007 99215 99306 99339 99511 99920 99007 99215 99306 99339 99512 99921 99007 99215 99306 99339 99512 99921 99008 99215 99310 99300 99339 99512 99921 99008 99215 99310 99400 99513 99907 99215 99310 99400 99513 99907 99216 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99555 99909 99911 99900 99215 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99551 99919 99009 99215 99311 99400 99550 99999 99111 99220 99331 99400 99550 99999 99111 99220 99331 99566 99999 99909 99111 99220 99331 99400 99550 99999 99900 99215 99311 99323 99331 99400 99550 99999 99909 99909 99909 99909 9 | | | | | | |
| 99047 99195 99289 99374 99487 99806 99048 99191 99290 99275 99488 99810 99048 9919 99200 99291 99375 99489 99811 99049 99200 99291 99376 99489 99811 99050 99201 99201 99376 99489 99811 99051 99201 99202 99377 99490 99814 99051 99202 9923 99377 99490 99814 99051 99203 99378 99496 99833 99052 99203 99204 99295 99380 99496 99833 99053 99205 99205 99205 99380 99496 99833 990554 99205 99206 99296 99381 99498 99488 99841 99056 99207 99382 99498 99881 99056 99207 99382 99498 99881 99056 99207 99382 99499 99881 99056 99208 99209 99384 99500 99894 99063 99208 99209 99384 99501 99887 99065 99208 99209 99386 99500 99889 99065 9920A 99300 99386 99503 99901 99065 9920A 99300 99386 99503 99901 99070 9920X 99301 99387 99505 99907 9920X 99301 99387 99505 99907 99071 09921 99302 99339 99364 99505 99907 99071 09921 99302 99339 99360 99389 99001 99071 09921 99302 99339 99360 99389 99001 99071 09921 99302 99339 99309 99505 99907 99077 99212 99304 99303 99309 99309 99309 99079 99071 09921 99304 99304 99309 9 | | | | | | |
| 99048 99199 99200 99291 99375 99488 99810 99049 99200 99291 99376 99489 99811 99050 99201 99202 99376 99480 99814 99051 99202 99293 99378 99495 99821 99052 99203 99293 99378 99495 99821 99052 99204 99295 99380 99497 99840 99053 99204 99295 99380 99497 99840 99055 99206 99296 99381 99499 99881 99056 99206 99297 99381 99499 99881 99058 99206 99297 99382 99499 99881 99058 99207 99298 99383 99500 99894 99060 99208 99299 99384 99500 99897 99060 99200 99300 99385 99500 99897 99060 99200 99300 99386 99500 99899 99070 99200 99300 99386 99500 99899 99070 99200 99301 99387 99504 99902 99071 99210 99303 99387 99504 99907 99072 99210 99303 99387 99504 99907 99072 99210 99303 99392 99506 99310 99074 99211 99302 99393 99391 99507 99913 99075 99212 99305 99394 99508 99913 99076 99213 99306 99393 99509 99913 99076 99214 99307 99306 99394 99509 99913 99077 99216 99308 99399 99399 99509 99914 99079 99216 99308 99399 99399 99509 99914 99079 99212 99306 99301 99395 99509 99914 99079 99212 99305 99394 99508 99913 99076 99213 99306 99397 99511 99920 99079 99078 99212 99308 99399 99399 99511 99920 99079 99079 99215 99308 99399 99511 99920 99079 99079 99215 99308 99399 99511 99920 99079 99078 99217 99310 99307 99316 99511 99920 99079 99078 99217 99310 99309 99399 99511 99920 99079 99079 99215 99310 99309 99399 99511 99920 99079 99215 99310 99309 99399 99511 99920 99099 99099999 99099 9909999 99099 990999 99099 99099999 99099 990999 99099 99 | | 99192 | | | 99486 | |
| 99049 99200 99201 99376 99483 99811 99050 99201 99292 99377 99490 99814 99051 99202 99377 99496 99814 99051 99202 99203 99378 99496 99831 99052 99203 99203 99204 99379 99496 99833 99503 99204 99295 99380 99497 99840 99840 99205 99205 99206 99381 99498 99841 99056 99205 99206 99381 99498 99881 99056 99207 99382 9449 99881 99058 99207 99382 9449 99881 99058 99207 99383 99500 99894 99500 99208 99209 99384 99501 99897 99060 99208 99209 99384 99501 99897 99060 99208 99209 99386 99500 99899 99399 99386 99503 99901 99070 99200 99300 99385 99503 99901 99070 99200 99300 99386 99503 99901 99070 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99301 99387 99506 99200 99301 99 | 99047 | 99195 | 99289 | 99374 | 99487 | 99806 |
| 99050 99201 99202 99377 99490 99814 99051 99202 99293 99378 99495 99813 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99058 99206 99297 99382 99499 99881 99058 99206 99297 99383 99500 99884 99059 99206 99297 99383 99500 99884 99050 99206 99299 99384 99501 99897 99060 99208 99299 99384 99501 99897 99060 99208 99299 99384 99501 99897 99060 99208 99300 99330 99335 99502 99889 99060 99208 99299 99384 99501 99897 99070 9920X 99301 9930 99386 99503 99901 99070 9920X 99301 9930 99386 99503 99901 99071 99210 99303 99302 99391 99506 99910 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99394 99508 99913 99076 99214 99307 99396 99396 99914 99077 99216 99306 99399 99396 99919 99079 99215 99306 99396 99396 99919 99079 99215 99308 99397 99511 99907 99078 99216 99308 99397 99511 99907 99079 99215 99308 99397 99511 99907 99078 99217 99310 99400 99399 99519 99919 99079 99215 99308 99397 99511 99907 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99929 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99079 99215 99308 99399 99551 99990 99089 99217 99311 99400 99551 99991 99078 99217 99313 99401 99551 99991 99079 99215 99318 99400 99551 99990 99089 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99319 99317 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99331 99401 99556 99990 99099 99214 99331 99404 99556 99990 99110 99226 99331 99446 99556 99999 99110 99236 99339 99344 99566 99999 99111 99236 99344 99446 99589 99999 99113 99244 99344 99448 99448 99660 | 99048 | 99199 | 99290 | 99375 | 99488 | 99810 |
| 99051 99202 99293 99378 99495 99821 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99056 99207 99298 99383 99500 99884 99056 99208 99299 99384 99501 99879 99060 99208 99299 99384 99501 99877 99063 99208 99299 99384 99501 99877 99065 9920A 99300 99386 99502 99889 99070 9920A 99300 99386 99503 99901 99071 09921 99302 99391 99505 99907 99071 09921 99302 99391 99505 99907 99074 99211 99304 99393 99506 99910 99075 99212 99305 99394 99506 99910 99076 99213 99306 99394 99506 99910 99077 99210 99307 99399 99507 99078 99214 99307 99399 99509 99914 99079 99215 99306 99399 99509 99914 99079 99216 99309 99399 99510 99919 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99079 99218 99311 99400 99513 99925 99080 99218 99311 99400 99539 99919 99080 99218 99311 99400 99539 99940 99080 99216 99315 99400 99552 99940 99099 99221 99315 99400 99554 99960 99099 99222 99317 99407 99555 99949 99099 99221 99318 99408 99557 99999 99091 99220 99317 99407 99555 99991 990910 99220 99317 99400 99555 99991 99010 99224 99331 99406 99555 99991 99100 99224 99331 99406 99555 99991 99101 99230 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99446 99566 99999 99114 99246 99344 99446 99593 99214 9 | 99049 | 99200 | 99291 | 99376 | 99489 | 99811 |
| 99051 99202 99293 99378 99495 99821 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99056 99207 99298 99383 99500 99884 99056 99208 99299 99384 99501 99879 99060 99208 99299 99384 99501 99877 99063 99208 99299 99384 99501 99877 99065 9920A 99300 99386 99502 99889 99070 9920A 99300 99386 99503 99901 99071 09921 99302 99391 99505 99907 99071 09921 99302 99391 99505 99907 99074 99211 99304 99393 99506 99910 99075 99212 99305 99394 99506 99910 99076 99213 99306 99394 99506 99910 99077 99210 99307 99399 99507 99078 99214 99307 99399 99509 99914 99079 99215 99306 99399 99509 99914 99079 99216 99309 99399 99510 99919 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99079 99218 99311 99400 99513 99925 99080 99218 99311 99400 99539 99919 99080 99218 99311 99400 99539 99940 99080 99216 99315 99400 99552 99940 99099 99221 99315 99400 99554 99960 99099 99222 99317 99407 99555 99949 99099 99221 99318 99408 99557 99999 99091 99220 99317 99407 99555 99991 990910 99220 99317 99400 99555 99991 99010 99224 99331 99406 99555 99991 99100 99224 99331 99406 99555 99991 99101 99230 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99432 99566 99999 99111 99231 99331 99446 99566 99999 99114 99246 99344 99446 99593 99214 9 | | | | | | |
| 99052 99203 99294 99295 99380 99497 99840 99054 99205 99286 99381 99498 99841 99056 99206 99297 99382 99499 99881 99058 99207 99298 99383 99500 99841 99060 99208 99299 99384 99501 9987 99063 99209 99384 99501 99897 99065 9920A 99300 99385 99503 99899 99076 9920A 99301 99387 99503 99899 99076 9920X 99301 99387 99504 99902 99071 09210 99302 99391 99505 99907 99072 99210 99303 99387 99506 99910 99074 99211 99304 99394 99506 99910 99075 99212 99305 9934 99508 99913 < | | | | | | |
| 99053 99204 9925 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99207 99288 99383 99500 99884 99063 99209 99300 99385 99501 99897 99063 9920A 99300 99386 99502 99899 99070 9920A 99300 99386 99503 99901 99071 09921 99301 99387 99504 99902 99071 09921 99302 99393 99505 99907 99072 99210 99303 99393 99505 99907 99074 99211 99304 99393 99507 99910 99075 99212 99305 99393 99507 99912 99076 99212 99305 99334 99508 99913 99078 99212 99307 9936 99510 9907 <t< td=""><td></td><td></td><td></td><td></td><td></td><td></td></t<> | | | | | | |
| 99056 99206 99297 99381 99498 99811 99056 99206 99297 99382 99499 99881 99058 99207 99298 99383 99500 99894 99060 99208 99299 99384 99501 99887 99063 99208 99299 99384 99501 99887 99065 9920A 99300 99385 99502 99899 99075 9920K 99301 99387 99505 99907 99071 09921 99302 99311 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99508 99914 99078 99214 99306 99395 99509 99914 99079 99215 99308 99397 99511 99920 99078 99216 99308 99397 99511 99920 99078 99216 99308 99397 99511 99920 99078 99216 99308 99399 99512 99079 99216 99308 99399 99512 99078 99216 99308 99399 99512 99079 99217 99310 99400 99513 99225 99080 99218 99311 99401 99514 99931 99081 99216 99319 99312 99401 99082 99216 99313 99401 99514 99931 99083 99216 99312 99402 99523 99940 99083 99216 99313 99403 99533 99942 99090 99215 99316 99404 99539 99519 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99555 99949 99091 99220 99317 99407 99555 99949 99091 99220 99317 99409 99554 99599 99091 99220 99317 99409 99554 99599 99091 99221 99318 99408 99558 99999 99104 99225 99324 9942 99559 99999 99104 99225 99324 99435 99446 99559 99999 99110 99236 99337 99447 99566 99999 99111 99236 99337 99447 99566 99999 99112 99238 9934 99447 99566 99999 99113 99244 99349 99447 99566 99999 99124 99245 99344 99344 99588 99999 9913 99246 99344 99447 99660 | | | | | | |
| 99056 99206 99297 99382 99499 99841 99058 99208 99298 99383 99500 99894 99060 99208 99299 99384 99501 99897 99063 99200 9930 99385 99502 99899 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99071 09921 99303 99393 99505 99907 99072 99210 99303 99393 99505 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99334 99508 99913 99076 99213 99306 99339 99509 99914 99078 99214 99307 99396 99510 99919 99078 99216 99309 99399 99512 99921 | 99053 | 99204 | 99295 | 99380 | 99497 | 99840 |
| 99058 99207 99298 99383 99500 99894 99060 99208 99299 99384 99501 99887 99063 99209 9930 99385 99502 99899 99065 9920A 99300 99386 99503 99901 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99075 99211 99304 99393 99507 99912 99076 99213 99306 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99309 99319 99507 99078 99216 99309 99309 99319 99500 99914 99079 99215 99308 99399 99512 99921 99070 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99311 99908 99082 9921F 99313 99402 99523 99940 99082 9921F 99313 99402 99530 99941 99089 99216 99317 99316 99404 99539 99940 99089 99216 99317 99316 99404 99539 99940 99089 99216 99317 99316 99404 99539 99940 99090 99215 99318 99316 99404 99539 99940 99090 99215 99316 99404 99555 99949 99091 99220 99317 99407 99552 99949 99091 99221 99318 99408 99553 99949 99091 99222 99321 99318 99408 99553 99949 99091 99223 99324 99324 99408 99553 99994 99091 99223 99324 99324 99408 99555 99949 99091 99223 99324 99324 99408 99555 99949 99091 99223 99324 99324 99408 99555 99996 9910 99224 99331 99408 99555 99996 9910 99225 99326 99325 99408 99555 99996 99110 99236 99325 99420 99558 99999 99110 99236 99326 99327 99426 99560 99999 99110 99236 99338 99349 99442 99560 99999 99110 99236 99338 99349 99442 99560 99999 99111 99236 99338 99349 99442 99560 99999 99112 99236 99338 99349 99442 99560 99999 99113 99234 99334 99344 99568 99999 99114 99236 99338 99344 99349 99560 99999 99115 99236 99338 99349 99442 99560 99999 99116 99236 99338 99344 99349 99560 99999 99119 99236 99338 99344 99349 99560 99999 99119 99236 99338 99349 99442 99560 99999 99130 99444 99546 99344 99544 99560 99999 99131 99246 99344 99344 99446 99593 99991 | 99054 | 99205 | 99296 | 99381 | 99498 | 99841 |
| 99060 99208 99299 99384 99501 9987 99063 99209 9930 99385 99502 99899 99070 9920A 99300 99387 99504 99901 99071 099210 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99910 99912 99076 99213 99305 99910 99912 99076 99213 99306 99395 99508 99913 99076 99213 99307 99396 99510 99912 99078 99214 99307 99396 99510 99919 99079 99215 99308 99399 99512 99921 99078 99216 99309 99319 99511 99921 9907 99217 </td <td>99056</td> <td>99206</td> <td>99297</td> <td>99382</td> <td>99499</td> <td>99881</td> | 99056 | 99206 | 99297 | 99382 | 99499 | 99881 |
| 99060 99208 99299 99384 99501 9987 99063 99209 9930 99385 99502 99899 99070 9920A 99300 99387 99504 99901 99071 099210 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99910 99912 99076 99213 99305 99910 99912 99076 99213 99306 99395 99508 99913 99076 99213 99307 99396 99510 99912 99078 99214 99307 99396 99510 99919 99079 99215 99308 99399 99512 99921 99078 99216 99309 99319 99511 99921 9907 99217 </td <td></td> <td>99207</td> <td></td> <td>99383</td> <td></td> <td></td> | | 99207 | | 99383 | | |
| 99063 99209 9930 99385 99502 99899 99065 9920A 99300 99385 99502 99899 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99392 99506 99910 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99395 99509 99914 99079 99215 99308 99397 99511 99920 99079 99215 99308 99399 99512 99921 99076 99217 99310 99400 99513 99922 99078 99218 99311 99400 99513 99925 99080 99218 99311 99401 99514 99931 99082 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99082 99217 99310 99402 99523 99940 99082 99217 99313 99402 99523 99940 99082 99217 99313 99403 99530 99941 99089 99216 99315 99404 99533 99942 99090 99215 99316 99400 99551 99940 99080 99218 99311 99402 99523 99940 99081 99219 99312 99402 99523 99940 99082 99217 99313 99403 99530 99941 99080 99218 99316 99404 99553 99940 99081 99219 99316 99400 99551 99940 99082 99216 99316 99400 99551 99964 99090 99215 99316 99400 99551 99940 99090 99215 99316 99400 99550 99941 99090 99215 99316 99406 99551 99949 99091 99220 99317 99407 99552 9949 99097 99221 99318 99409 99554 99959 99097 99221 99318 99409 99554 99960 99077 99221 99318 99409 99554 99960 99099 99222 99321 99400 99554 99960 99099 99222 99321 99409 99554 99960 99099 99222 99321 99409 99554 99960 99091 99220 99317 99407 99552 9949 99091 99220 99317 99407 99552 9949 99091 99220 99317 99407 99554 99999999999999999999999999999999 | | | | | | |
| 99065 9920A 99300 99386 99503 99901 99070 9920K 99301 99387 9950A 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99333 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99926 99078 99218 99311 99400 99513 99925 99080 99218 99311 99400 99513 99925 99080 99218 99311 99400 99513 99925 99082 9921F 99313 99402 99523 9940 99082 9921F 99313 99403 99530 99941 99089 99099 99212 99315 99404 99539 99942 99099 99212 99316 99309 99404 99539 99949 99099 99215 99316 99309 99404 99539 99949 99099 99215 99316 99404 99539 99949 99099 99215 99316 99404 99539 99949 99099 99215 99316 99404 99539 99949 99099 99215 99316 99404 99539 99949 99099 99215 99316 99404 99539 99949 99091 99215 99316 99404 99539 99949 99099 99215 99316 99404 99539 99949 99091 99215 99316 99406 99551 99949 99099 99215 99316 99408 99553 99949 99099 99215 99316 99408 99553 99949 99099 99219 99319 99319 99409 99554 99960 99099 99220 99317 99409 99554 99960 99099 99220 99321 99409 99554 99960 99099 99220 99321 99409 99556 99969 99010 99224 99323 99322 9940A 99555 99961 99101 99226 99325 99324 99412 99557 99970 99102 99226 99325 99326 99429 99559 99999 99101 99226 99325 99326 99429 99559 99999 99110 99230 99327 99426 99560 99999 99110 99230 99331 99326 99431 99560 99999 99110 99230 99331 99332 99440 99560 99999 99111 99231 99336 99431 99566 99999 99111 99231 99336 99431 99566 99999 99112 99234 99331 99434 99438 99566 99999 99112 99234 99331 99444 99568 99999 99124 99349 99344 99446 99569 99999 99124 99349 99349 99444 99569 99999 99124 99349 99344 99446 99569 99999 99124 99349 99349 99444 99569 99999 99124 99349 99349 99444 99569 99999 99124 99349 99444 99344 99569 99999 99124 99344 99344 99446 99588 99999 99124 99344 99344 99448 99660 | | | | | | |
| 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99925 99081 99218 99311 99401 99514 99931 99082 99218 99311 99401 99514 99931 99082 9921F 99312 99402 99523 99940 99089 99216 99315 99404 99539 99542 99099 99215 99316 99404 99539 99941 99099 99215 99316 99400 99551 99940 99089 99216 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99599 99099 99222 99321 99408 99553 99599 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99408 99553 99959 99099 99221 99318 99408 99553 99959 99099 99221 99318 99408 99553 99959 99099 99222 99321 99408 99553 99960 9901 99220 99317 99407 99552 99949 9901 99220 99317 99409 99554 99960 9901 99220 99317 99409 99554 99960 9901 99220 99317 99409 99554 99960 9901 99220 99319 99409 99554 99960 9901 99220 99319 99409 99554 99960 9901 99220 99321 99409 99554 99960 9901 99220 99321 99409 99554 99960 9901 99220 99321 99326 99409 99559 99999 9910 99220 99321 99409 99559 99999 9910 99221 99336 99409 99559 99999 9910 99221 99336 99449 99559 99999 9910 99221 99336 99340 99559 99999 99110 99230 99327 99426 99560 99999 99110 99230 99337 99426 99560 99999 99110 99230 99337 99446 99566 99999 99110 99230 99337 99441 99568 99999 99110 99230 99337 99441 99568 99999 99110 99230 99339 99337 99444 99569 99999 99110 99230 99339 99337 99444 99569 99999 99111 99236 99339 99344 99446 99569 99999 99112 99236 99339 99344 99446 99569 99999 99124 99244 99340 99448 99560 99999 99124 99245 99343 99447 99600 | | | | | | |
| 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99508 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99511 99920 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99079 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99218 99311 99401 99523 99940 99081 99219 99312 99402 99523 99941 99089 99216 99315 99403 99539 99942 99089 99216 | 99065 | 9920A | 99300 | 99386 | 99503 | 99901 |
| 99072 99210 99303 99392 99506 99910 99074 99211 99304 99333 99507 99912 99075 99212 99306 99394 99508 99913 99076 99213 99306 99395 99500 99914 99078 99214 99307 99396 99510 99919 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99511 99920 99078 99216 99309 99319 99511 99921 99078 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 9982 99216 99315 99402 99530 99941 | 99070 | 9920X | 99301 | 99387 | 99504 | 99902 |
| 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99078 99213 99306 99395 99510 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99512 99921 99078 99216 99300 99313 99921 99078 99216 99300 99313 99921 99079 99217 99310 99400 99513 99921 9907 99217 99310 99401 99514 99931 99080 99218 99311 99401 99514 99931 99082 99216 99315 99402 9953 99942 99091 99215 99316 99406 99551 99943 99091 99220 99317 </td <td>99071</td> <td>09921</td> <td>99302</td> <td>99391</td> <td>99505</td> <td>99907</td> | 99071 | 09921 | 99302 | 99391 | 99505 | 99907 |
| 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99078 99213 99306 99395 99510 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99512 99921 99078 99216 99300 99313 99921 99078 99216 99300 99313 99921 99079 99217 99310 99400 99513 99921 9907 99217 99310 99401 99514 99931 99080 99218 99311 99401 99514 99931 99082 99216 99315 99402 9953 99942 99091 99215 99316 99406 99551 99943 99091 99220 99317 </td <td>99072</td> <td>99210</td> <td>99303</td> <td>99392</td> <td>99506</td> <td>99910</td> | 99072 | 99210 | 99303 | 99392 | 99506 | 99910 |
| 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 9921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99081 99219 99312 99402 99523 99940 99082 99216 99313 99403 99530 99941 99089 99216 99315 99404 99539 99942 99090 99215 99316 99406 99551 99943 99090 99215 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 | | | | | | |
| 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99339 99512 99921 99078 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 99215 99316 99404 99539 99943 99001 99220 99317 99407 99551 99949 99007 99215 99318 99408 99551 99949 99097 99221 99318 99408 99553 99959 | | | | | | |
| 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99076 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 9931 99081 99219 99312 99402 99533 99940 99082 99216 99313 99403 99530 99941 99089 99216 99315 99404 99539 99942 99090 99215 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99409 99554 9960 99057 99221 9931 99409 99554 9966 <tr< td=""><td></td><td></td><td></td><td></td><td></td><td></td></tr<> | | | | | | |
| 99079 99215 99308 99397 99511 99920 9907B 99216 99309 99319 99512 99921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99408 99554 99960 9957 99223 99322 99408 99555 99961 | 99076 | 99213 | 99306 | 99395 | 99509 | 99914 |
| 9907B 99216 99309 99399 99512 99921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99408 99553 99959 99097 99221 99321 99409 99554 99960 99057 99223 99321 99409 99554 99960 99057 99223 99324 99419 99556 99961 | 99078 | 99214 | 99307 | 99396 | 99510 | 99919 |
| 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 9922O 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99407 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 99409 99554 99960 99057 99223 99322 99409 99555 99961 99100 99224 99323 99411 99557 99970 | 99079 | 99215 | 99308 | 99397 | 99511 | 99920 |
| 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 9922O 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99407 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 99409 99554 99960 99057 99223 99322 99409 99555 99961 99100 99224 99323 99411 99557 99970 | 9907B | 99216 | 99309 | 99399 | 99512 | 99921 |
| 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 9943 99091 99220 99317 99407 99552 9949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99408 99553 99959 99097 99221 99318 99408 99553 99959 99099 99222 99321 99408 99554 99960 99007 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 < | 9907F | | 99310 | 99400 | 99513 | 99925 |
| 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99961 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9988 99104 99227 99326 99420 99558 99989 99110 99230 99327 99426 99560 99990 | | | | | | |
| 99082 9921F 99313 99403 99530 9941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 9960 990ST 99223 99322 9940A 99555 9961 99100 99224 99323 99411 99556 9996 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99420 99558 9989 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 | | | | | | |
| 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99999 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 | | | | | | |
| 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99999 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 | 99082 | 9921F | 99313 | 99403 | 99530 | 99941 |
| 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99332 99331 99432 99562 99992 99113 99233 99332 99433 99564 99994 99115 99234 99333 99435 99564 99994 | 99089 | 9921G | 99315 | 99404 | 99539 | 99942 |
| 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 9905T 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 <t< td=""><td>99090</td><td>9921S</td><td>99316</td><td>99406</td><td>99551</td><td>99943</td></t<> | 99090 | 9921S | 99316 | 99406 | 99551 | 99943 |
| 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 9905T 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 <t< td=""><td>99091</td><td>99220</td><td>99317</td><td>99407</td><td>99552</td><td>99949</td></t<> | 99091 | 99220 | 99317 | 99407 | 99552 | 99949 |
| 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 9991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 9994 99116 99235 99344 99436 99565 99995 99119 99236 99335 99438 99566 99996 <tr< td=""><td></td><td></td><td></td><td></td><td></td><td></td></tr<> | | | | | | |
| 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 9991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 < | | | | | | |
| 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99344 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99999 | | | | | | |
| 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 | | | | | | |
| 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 < | 99100 | | 99323 | 99411 | 99556 | 99968 |
| 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V | 99101 | 99225 | 99324 | 99412 | 99557 | 99970 |
| 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V | 99102 | 99226 | 99325 | 99420 | 99558 | 99989 |
| 99110 99230 99327 9942G 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 9931 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 | | | 99326 | | 99559 | |
| 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99933 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99344 99448 99600 | | | | | | |
| 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99113 | 99233 | 99332 | 99433 | 99563 | 99993 |
| 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99115 | 99234 | 99333 | 99435 | 99564 | 99994 |
| 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99116 | 99235 | 99334 | 99436 | 99565 | 99995 |
| 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | 99236 | | | 99566 | |
| 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99714 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | 99241 | 99339 | 99442 | 99569 | 99999 |
| 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99124 | 99242 | 99340 | 99443 | 99580 | 9999G |
| 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99125 | 99243 | 99341 | 99444 | 99588 | 9999V |
| 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 09913 | 99244 | 99342 | 99446 | 99593 | 99Z14 |
| 09914 99246 99344 99448 99601 | | | | | | |
| 99140 99345 99449 99602 | | | | | | |
| | 99140 | 99248 | 99345 | 99449 | 99602 | |



# Appendix A Healthcare utilization measures

| 86140 | 86141 |
|-------|-------|

#### Number of serum creatinine tests

| italiibei oi seraili a | cutiline tests |
|------------------------|----------------|
| CPT | |
| 80048 | 80054 |
| 80049 | 80069 |
| 80053 | 82565 |

#### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| ntestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality Disorders, And Other Nonpsychotic Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.800, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.283, F16.288, F16.980, F16.983, F16.983, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.950, F19.951, F19.96, F19.282, F19.991, F19.982, F19.993, F19.94, F19.950, F19.951, F19.96, F19.282, F19.991, F19.982, F19.994, F19.950, F19.951, F19.96, F19.282, F19.991, F19.982, F19.994, F19.950, F19.951, F19.96, F19.282, F19.991, F19.982, F19.994, F19.950, F19.951, F19.96, F19.282, F19.991, F19.982, F19.994, F19.950, F19.951, F19.96, F19.282, F19.991, F19.994, F19.995, F19.950, F19.951, F19.96, F19.282, F19.991, F19.994, F19.995, F19.950, F19.951, F19.96, F19.282, F19.994, F19.995, F | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-<br>G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | J30-J39 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36<br>(excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | S81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

Osteoporosis

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| 80702 | Multiple fractures of ribs, bilateral, initial encounter for | Closed fracture of two ribs |
|---|---|---|
| 80703 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of three ribs |
| 80703 | Multiple fractures of ribs, left side, initial encounter for | Closed fracture of three ribs |
| | closed fracture | |
| 80703 | · · | Closed fracture of three ribs |
| 80703 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of three ribs |
| 80704 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of four ribs |
| 80704 | Multiple fractures of ribs, left side, initial encounter for closed fracture | Closed fracture of four ribs |
| 80704 | Multiple fractures of ribs, bilateral, initial encounter for | Closed fracture of four ribs |
| 80704 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of four ribs |
| 80705 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of five ribs |
| 80705 | Multiple fractures of ribs, left side, initial encounter for | Closed fracture of five ribs |
| 80705 | Multiple fractures of ribs, bilateral, initial encounter for | Closed fracture of five ribs |
| 80705 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of five ribs |
| 80706 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of six ribs |
| 80706 | Multiple fractures of ribs, left side, initial encounter for | Closed fracture of six ribs |
| 80706 | Multiple fractures of ribs, bilateral, initial encounter for | Closed fracture of six ribs |
| 80706 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of six ribs |
| 80707 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of seven ribs |
| 80707 | Multiple fractures of ribs, left side, initial encounter for closed fracture | Closed fracture of seven ribs |
| 80707 | Multiple fractures of ribs, bilateral, initial encounter for closed fracture | Closed fracture of seven ribs |
| 80707 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of seven ribs |
| 80708 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of eight or more ribs |
| 80708 | Multiple fractures of ribs, left side, initial encounter for closed fracture | Closed fracture of eight or more ribs |
| 80708 | Multiple fractures of ribs, bilateral, initial encounter for closed fracture | Closed fracture of eight or more ribs |
| 80708 | Multiple fractures of ribs, unspecified side, initial encounter | Closed fracture of eight or more ribs |
| 80709 | Multiple fractures of ribs, right side, initial encounter for | Closed fracture of multiple ribs, unspecified |
| 80709 | Multiple fractures of ribs, left side, initial encounter for | Closed fracture of multiple ribs, unspecified |
| 80709 | Multiple fractures of ribs, bilateral, initial encounter for | Closed fracture of multiple ribs, unspecified |
| 80710 | Fracture of one rib, unspecified side, initial encounter for open fracture | Open fracture of rib(s), unspecified |
| 80711 | Fracture of one rib, right side, initial encounter for open | Open fracture of one rib |
| 80711 | Fracture of one rib, left side, initial encounter for open fracture | Open fracture of one rib |
| | 80703<br>80703<br>80703<br>80703<br>80703<br>80704<br>80704<br>80704<br>80704<br>80705<br>80705<br>80705<br>80705<br>80706<br>80706<br>80706<br>80706<br>80707<br>80709<br>80710<br>80711 | dosed fracture 80703 Multiple fractures of ribs, right side, initial encounter for dosed fracture 80703 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80703 Multiple fractures of ribs, bilateral, initial encounter for dosed fracture 80703 Multiple fractures of ribs, unspecified side, initial encounter for dosed fracture 80704 Multiple fractures of ribs, right side, initial encounter for dosed fracture 80704 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80704 Multiple fractures of ribs, bilateral, initial encounter for dosed fracture 80704 Multiple fractures of ribs, unspecified side, initial encounter for dosed fracture 80705 Multiple fractures of ribs, right side, initial encounter for dosed fracture 80705 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80705 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80705 Multiple fractures of ribs, unspecified side, initial encounter for dosed fracture 80706 Multiple fractures of ribs, unspecified side, initial encounter for dosed fracture 80706 Multiple fractures of ribs, right side, initial encounter for dosed fracture 80706 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80706 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80706 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80707 Multiple fractures of ribs, unspecified side, initial encounter for dosed fracture 80708 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80707 Multiple fractures of ribs, right side, initial encounter for dosed fracture 80708 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80708 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80708 Multiple fractures of ribs, left side, initial encounter for dosed fracture 80709 Multiple fractures of ribs, left side, initial encounter for dosed fracture |


# Appendix A Frailty markers


# Falls


# Appendix A Frailty markers

## Combined Comorbidity Score for Claims Data

Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her O. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


# Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

# Appendix A Comedications

## Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

# Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| Anti epitepite non mood stabilizers | |
|-------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

## Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

## Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

# Selective serotonin reuptake inhibitor

| NDC Generic Name | |
|---------------------------|-----------------------------------------|
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

# Tricyclic antidepressants

| NDC Generic Name | |
|------------------------------------|--------------------------------|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL |
| AMOXAPINE | DOXEPIN HCL |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL |

# Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

# Appendix A Comedications

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

### Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM,PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM,PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM,PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| Antiplatelet agents | |
|---|---|
| NDC Generic Name | |
| ABCIXIMAB | CILOSTAZOL |
| ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | VORAPAXAR SULFATE |
| NDC Brand Name | |
| ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

## Angiotensin II Receptor Blockers

| NDC Generic Name | |
|---|---|
| ALISKIREN/VALSARTAN | LOSARTAN POTASSIUM |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE/VALSARTAN | OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZID |
| AZILSARTAN MEDOXOMIL | OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE | TELMISARTAN |
| CANDESARTAN CILEXETIL | TELMISARTAN/AMLODIPINE BESYLATE |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE | TELMISARTAN/HYDROCHLOROTHIAZIDE |
| IRBESARTAN | VALSARTAN |

| IRBESARTAN/HYDROCHLOROTHIAZIDE | VALSARTAN/HYDROCHLOROTHIAZIDE |
|--------------------------------|--------------------------------|
| NDC Brand Name | · |
| AMLODIPINE-VALSARTAN | EXFORGE HCT |
| ATACAND | HYZAAR |
| ATACAND HCT | IRBESARTAN |
| AVALIDE | IRBESARTAN-HYDROCHLOROTHIAZIDE |
| AVAPRO | LOSARTAN POTASSIUM |
| AZOR | LOSARTAN-HYDROCHLOROTHIAZIDE |
| BENICAR | MICARDIS |
| BENICAR HCT | MICARDIS HCT |
| CANDESARTAN CILEXETIL | TELMISARTAN |
| CANDESARTAN-HYDROCHLOROTHIAZID | TELMISARTAN-AMLODIPINE |
| COZAAR | TELMISARTAN-HYDROCHLOROTHIAZID |
| DIOVAN | TRIBENZOR |
| DIOVAN HCT | TWYNSTA |
| EDARBI | VALSARTAN |
| EDARBYCLOR | VALSARTAN-HYDROCHLOROTHIAZIDE |
| EXFORGE | VALTURNA |

| Angiotensin Converting Enzyme inhibitors | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | LISINOPRIL |
| BENAZEPRIL HCL | LISINOPRIL/HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE | MOEXIPRIL HCL |
| CAPTOPRIL | MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | PERINDOPRIL ERBUMINE |
| ENALAPRIL MALEATE | QUINAPRIL HCL |
| ENALAPRIL MALEATE/FELODIPINE | QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE | RAMIPRIL |
| ENALAPRILAT DIHYDRATE | TRANDOLAPRIL |
| FOSINOPRIL SODIUM | TRANDOLAPRIL/VERAPAMIL HCL |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ACCUPRIL | LOTREL |
| ACCURETIC | LYTENSOPRIL |
| ACEON | LYTENSOPRIL-90 |
| ALTACE | MAVIK |
| AMLODIPINE BESYLATE-BENAZEPRIL | MOEXIPRIL HCL |
| BENAZEPRIL HCL | MOEXIPRIL-HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL-HCTZ | MONOPRIL |
| BENAZEPRIL-HYDROCHLOROTHIAZIDE | MONOPRIL HCT |
| CAPOTEN | PERINDOPRIL ERBUMINE |
| CAPOZIDE | PRINIVIL |
| CAPTOPRIL | PRINZIDE |
| CAPTOPRIL-HYDROCHLOROTHIAZIDE | QUINAPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | QUINAPRIL HCL |
| ENALAPRIL MALEATE | QUINAPRIL-HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE-HCTZ | QUINARETIC |
| ENALAPRIL MALEATE/HCTZ | RAMIPRIL |
| ENALAPRIL-HYDROCHLOROTHIAZIDE | TARKA |
| ENALAPRILAT | TRANDOLAPRIL |
| EPANED | TRANDOLAPRIL-VERAPAMIL |
| FOSINOPRIL SODIUM | UNIRETIC |
| FOSINOPRIL-HYDROCHLOROTHIAZIDE | UNIVASC |
| LEXXEL | VASERETIC |
| LISINOPRIL | VASOTEC |
| LISINOPRIL-HCTZ | VASOTEC I.V. |
| LISINOPRIL-HYDROCHLOROTHIAZIDE | ZESTORETIC |
| LOTENSIN | ZESTRIL |
| LOTENSIN HCT | |

#### Beta blockers

| Deta Blockers | |
|-------------------------|------------------------------------------|
| NDC Generic Name | |
| ACEBUTOLOL HCL | ESMOLOL HCL |
| ATENOLOL | LABETALOL HCL |
| ATENOLOL/CHLORTHALIDONE | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| BISOPROLOL FUMARATE | METOPROLOL TARTRATE |

| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE | METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
|---|---|
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE | NEBIVOLOL HCL |
| CARTEOLOL HCL | SOTALOL HCL |
| CARVEDILOL | TIMOLOL |
| CARVEDILOL PHOSPHATE | TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE | TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF | TIMOLOL MALEATE/PF |
| NDC Brand Name | |
| ACEBUTOLOL HCL | ISTALOL |
| ATENOLOL | KERLONE |
| ATENOLOL W/CHLORTHALIDONE | LABETALOL HCL |
| ATENOLOL-CHLORTHALIDONE | LOPRESSOR |
| BETAPACE | LOPRESSOR HCT |
| BETAPACE AF | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL TARTRATE |
| BETIMOL | METOPROLOL-HYDROCHLOROTHIAZIDE |
| BETOPTIC | NORMODYNE |
| BETOPTIC S | OCUPRESS |
| BISOPROLOL FUMARATE | SECTRAL |
| BISOPROLOL FUMARATE-HCTZ | SENORMIN |
| BISOPROLOL FUMARATE/HCTZ | SORINE |
| BISOPROLOL-HYDROCHLOROTHIAZIDE | SOTALOL |
| BLOCADREN | SOTALOL AF |
| BREVIBLOC | SOTALOL HCL |
| BYSTOLIC | TENORETIC 100 |
| CARTEOLOL HCL | TENORETIC 50 |
| CARTROL | TENORMIN |
| CARVEDILOL | TENORMIN CALENDAR PAK |
| COMBIGAN | TIMOLIDE |
| COREG | TIMOLOL MALEATE |
| COREG CR | TIMOPTIC |
| COSOPT | TIMOPTIC OCUDOSE |
| COSOPT PF | TIMOPTIC-XE |
| DORZOLAMIDE-TIMOLOL | TOPROL XL |
| DUTOPROL | TRANDATE |
| ESMOLOL HCL | ZEBETA |
| HYPERTENSOLOL | ZIAC |

# Calcium channel blockers

| Calcium channel blockers | |
|---|---|
| HCPCS | |
| C9248 | |
| NDC Generic Name | |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE | BEPRIDIL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE | CLEVIDIPINE BUTYRATE |
| AMLODIPINE BESYLATE | DILTIAZEM HCL |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | DILTIAZEM MALATE |
| AMLODIPINE BESYLATE/VALSARTAN | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |

# Appendix A Comedications

| CARDIZEM CD | NYMALIZE |
|-------------------|------------------------|
| CARDIZEM LA | PLENDIL |
| CARDIZEM SR | POSICOR |
| CARTIA XT | PROCARDIA |
| CLEVIPREX | PROCARDIA XL |
| COVERA-HS | SULAR |
| DILACOR XR | TARKA |
| DILT-CD | TAZTIA XT |
| DILT-XR | TEKAMLO |
| DILTIA XT | TELMISARTAN-AMLODIPINE |
| DILTIAZEM 24HR CD | TIAMATE |
| DILTIAZEM 24HR ER | TIAZAC |
| DILTIAZEM ER | TRANDOLAPRIL-VERAPAMIL |
| DILTIAZEM HCL | TRIBENZOR |
| DILTIAZEM HCL-NS | TWYNSTA |
| DILTIAZEM XR | VASCOR |
| DILTIAZEM-D5W | VERAPAMIL ER |
| DILTZAC ER | VERAPAMIL ER PM |
| DYNACIRC | VERAPAMIL HCL |
| DYNACIRC CR | VERAPAMIL SR |
| EXFORGE | VERELAN |
| EXFORGE HCT | VERELAN PM |
| FELODIPINE ER | |

## Diuretics

| NDC Generic Name | |
|-----------------------------------|---------------------|
| AMILORIDE HCL | HYDROCHLOROTHIAZIDE |
| AMILORIDE HCL/HYDROCHLOROTHIAZIDE | HYDROFLUMETHIAZIDE |
| BENDROFLUMETHIAZIDE | INDAPAMIDE |
| BUMETANIDE | METHYCLOTHIAZIDE |
| CHLOROTHIAZIDE | METOLAZONE |
| CHLORTHALIDONE | POLYTHIAZIDE |
| EPLERENONE | SPIRONOLACTONE |
| ETHACRYNATE SODIUM | TORSEMIDE |
| ETHACRYNIC ACID | TRIAMTERENE |
| FUROSEMIDE | TRICHLORMETHIAZIDE |

# Nitrates

| Nitrates | |
|---|---|
| NDC Generic Name | NDC Generic Name |
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL | NITROGLYCERIN/DEXTROSE 5 % IN WATER |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |
| DILATRATE-SR | NITROCINE |
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 | NITROMIST |
| ISOREX-2.5 | NITRONAL |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |

# Appendix A Comedications

| ISOTRATE ER | NITROSTAT IV |
|--------------------------|-----------------|
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| Lipid lowering drugs | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | METHYLTETRAHYDROFOLATE GLUCOSAMINE/NIACINAMIDE/CUPRIC &ZN OX |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA | NIACIN |
| ATORVASTATIN CALCIUM | NIACIN (INOSITOL NIACINATE) |
| BETA-CAROTENE(A) W-C & E/NIACINAMIDE/VIT B2/LUT/MIN/GLU-ONE | NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| CERAMIDES 1,3,6-11/NIACINAMIDE | NIACIN/LOVASTATIN |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID | NIACIN/SIMVASTATIN |
| CHOLESTYRAMINE | NIACINAMIDE |
| CHOLESTYRAMINE (WITH SUGAR) | NIACINAMIDE ASCORBATE |
| CHOLESTYRAMINE/ASPARTAME | NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| COLESEVELAM HCL | NIACINAMIDE/RIBOFLAVIN/BETA-CAROTENE(A) W-C & E/MINERALS |
| COLESTIPOL HCL | NIACINAMIDE/VIT B6/VIT C/FA/COPPER/MG CIT/ZN GLUC/ALIP ACID |
| EZETIMIBE | PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| EZETIMIBE/ATORVASTATIN CALCIUM | PITAVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN | POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| FENOFIBRATE | PRAVASTATIN SODIUM |
| FENOFIBRATE NANOCRYSTALLIZED | ROSUVASTATIN CALCIUM |
| FENOFIBRATE,MICRONIZED | SIMVASTATIN |
| FLUVASTATIN SODIUM | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| FOLIC ACID/NIACINAMIDE/ZINC | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| GEMFIBROZIL | THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| INOSITOL NIACINATE | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |
| | <del>-</del> |

### Non-insulin diabetes medications

| Non-insulin diabetes inedications | |
|--------------------------------------|-------------------------------------|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL | PIOGLITAZONE HCL/METFORMIN HCL |
| CANAGLIFLOZIN/METFORMIN HCL | REPAGLINIDE |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |

| GLYBURIDE | SAXAGLIPTIN HCL |
|---|---|
| GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | TOLAZAMIDE |
| METFORMIN/CAFFEINE/AMINO ACIDS#7/HERBAL COMB#125/CHOLINE BIT | TOLBUTAMIDE |
| NDC Brand Name | |
| ACARBOSE | ICN-TOLAM |
| ACETOHEXAMIDE | INSULASE |
| ACTOPLUS MET | INVOKAMET |
| ACTOPLUS MET XR | JANUMET |
| ACTOS | JANUMET XR |
| AMARYL | JANUVIA |
| APPFORMIN | JENTADUETO |
| APPFORMIN-D | JUVISYNC |
| AVANDAMET | KAZANO |
| AVANDARYL | KOMBIGLYZE XR |
| AVANDIA | METAGLIP |
| CHLORABETIC 250 | METFORMIN HCL |
| CHLORPROPAMIDE | METFORMIN HCL ER |
| DIABETA | MICRONASE |
| DIABINESE | NATEGLINIDE |
| DIBATROL | NESINA |
| DUETACT | ONGLYZA |
| DYMELOR | ORIBETIC |
| FORTAMET | ORINASE |
| GLIMEPIRIDE | OSENI |
| GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCAMIDE | PRANDIN |
| GLUCOPHAGE | PRECOSE |
| GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOTROL | RIOMET |
| GLUCOTROL XL | RONASE |
| GLUCOVANCE | SK-TOLBUTAMIDE |
| GLUMETZA | STARLIX |
| GLYBURIDE | TOLAMIDE |
| GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| GLYCRON | TOLINASE |
| GLYNASE | TRADJENTA |
| GLYSET | |

# Insulin


# Appendix A Comedications

| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
|-----------------------------|--------------------------------|
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| HUMALOG MIX 50/50 | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | |

## Antidepressants

| HCPCS | |
|---|---|
| J1320 | |
| NDC Generic Name | |
| AMITRIPTYLINE HCL | IMIPRAMINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEVOMILNACIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT, MISC. COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE | VORTIOXETINE HYDROBROMIDE |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |

| AMONAPINE MINTAZAPHE ANYDROUS ANAPETAMIN PREDITAMONE PREDITAMONE NOFERAMIN NEFACOONE HCI NOFERAMIN NEFACOONE HCI NOFERAMIN NOFERAMIN NOFERAMIN NOFERAMIN NORTRIPTYLINE HCI OLANZARMIN HCI OLANZARMIN HCI SENDERICH PAMELOR BUDEPRION SR BUDEPRION SR PAMELOR BUDEPRION SR PARKIC R BUDEPRION SR PARKIC R BUDEPRION NL PARKIC R BUDEPRION NL PARKIC R BUDEPRION NL PARKIC R BUDEPRION NL PERTERIP BUDEPRION NL PERTERIP BUDEPRION HCI ER PERTERIP BUDEVER HCI ER BUDEPRION HCI ER BUDEPR | AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
|---|---|---|
| AMAFABIL APRIEZIM NARONE APPRITAMONE NOBERAMI NO | · | |
| NEFACOONE INC. | | |
| MORFRANII | | |
| APSENDIN MORTAMINE HU. APSENDIN MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO M. BR | | |
| ASENDIN | | |
| AVENTYL HCL OLANAZARIK-FLUXXETINE HCL BRISTELIX BRISTELIX BRISTELIX DEFPROR N. BRISTELIX PARKICR BLUDEPRON X. PEXEVA PEXEVA PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. BLUPROPHON X. PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. PROSE BLUPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUD X. BLUDEPROPHON X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDR | | |
| SINTELLIX OLEFTO & R | | |
| RRISDELLE PAMELOR PARCETINE H.C. PERPERBAN PARCETINE H.C. PERPERBAN PERPENBAN PERPENBA | | |
| BRUDEPRION SR | | |
| PAXIL PAXI | | |
| BURDEDAN PAXIL CR | | |
| BURDOPION H.C. PERTER | | |
| BURDOPION HCL ER BURDOPION HCL SR BURDOPION SC PEXEVA BURDOPION SC PEXEVA BURDOPION SC PERCENA PRISTIQ ER BURDOPION SC PROTECT | | |
| BURDOPION HCL SR | | |
| PURPOPION XL | | |
| CELEXA PROTREPTYLINE HCL CHTALOPRAM PROZAC CITALOPRAM HRR PROZAC REHIVE DESIPRAM DESVENILATANIE FROM DESVENILATANIE SERTRALINE HCL TRAVIL 10-2 | | |
| CHIORDIAZEPOXIDE-AMITRIPTYUNE PROZAC CITALOPRAM PROZAC CWERKLY PRUDOXIN CYMBALTA Q.E. L DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RE-LUVE DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FUMARATE ER SARAFEM SELFEMRA DOKERIH HCL SENTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE PROLOXE PVILL 10 SERZONE FVILL 10 SERZONE FVILL 25 SINEQUAN SK-PAMITRIPTYUNE SK-PAMITRIPTY | | |
| CITALOPRAM HBR PROZAC C TITALOPRAM HBR PROZAC WEEKLY CICMIPPAMINE HCL PRUDOWN CYMBALTA Q.E.L PRUDOWN CICMIPPAMINE HCL PRUDOWN CESTINAL Q.E.L PRUDOWN DESIPHARMINE HCL RAPPILUX DESIPHARMINE HCL REHVE DESIPHARMINE HCL REHVE DESIVENLAFAXINE ER REMERON DESVENLAFAXINE FUMARATE ER SARAFEM DESVENLAFAXINE FUMARATE ER SELFEMRA DOXEPIN HCL SENTROXATINE DOXEPIN HCL SENTROXATINE DULONEITIEN HCL SERTRALINE SERTRALINE SERTRALIN | | |
| PROZAC WEEKLY | | |
| PRIDOXIN | | |
| CYMBALTA | | |
| DECONIL RAPIFLUX DESSIPRAMINE HCL RE-UVE DESSIPRAMINE HCL RE-UVE REMERON DESSIPRAMINE FUNARATE ER REMERON DESSURLAFAXINE FUMARATE ER SELFEMRA DOXEDIH HCL SERTROWATINE DOULOXETINE HCL SERTROWATINE SELFEMRA SILENOR E-VILL 100 SILENOR E-VILL 100 SILENOR E-VILL 55 SINEQUAN SERVALISO SK-AMITIRIPTYLINE E-VILL 50 SK-AMITIRIPTYLINE E-VILL 75 SK-PAMINE STABANIL STEFEXOR STABANIL SURMONTIL E-FEXOR SURMONTIL E-BAYL SURMONTIL E-MITRIP TOFRANIL-PM FINOVIL STABANIL SOTTALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-5 TRIAVIL 2-6 TRIAVIL 3-6 ELUXOKANINE MALEATE TRIAVIL 4-10 FILIOXETINE HCL TRIAVIL 4-10 FILIOXETINE HCL FILIOXETINE HCL TRIAVIL 4-10 TRIAVIL 4-10 FILIOXETINE HCL FILIOXETINE HCL TRIAVIL 4-10 TRIAVIL 4-10 FILIOXETINE HCL TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-10 FILIOXETINE HCL TRIAVIL 4-10 T | | |
| DESIPRAMINE HCL DESVENLAFAXINE FUMARATE ER DESVENLAFAXINE MCL DULOXETINE HCL SERTROLATINE SERTROLATINE SERTROLATION SERTROLATINE SERTROLATION | | · |
| DESVENLAFAXINE ER DESVENLAFAXINE FUMARATE ER DESYREL SELFEMRA DOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SILENOR STABANIL SEFEXOR STABANIL SEFEXOR STABANIL SERVILL STABA | | |
| DESVENLAFAXINE FUMARATE ER SERFEMRA DOSYPRIL SELFWRA DOSYPRIL SELFWRA DOLOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE SIMEOUAN SERTRALINE SERTRALI | | |
| DESYREL DESYREL SELFEMRA DOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE SERTRALINE HCL SERTRALINE SERTRAL | | |
| DOUCRPIN HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SILENOR SEAMITRIPTYLINE EVILL 75 SEPRAMINE SEFEXOR STABANIL SEFEXOR STABANIL SUMMONTIL SELAVIL SYMBYAX SILENOR SILENOR STABANIL SYMBYAX SILENOR STABANIL SELAVIL SELAVIL SELAV | | |
| DULOXETINE HCL SERTABLINE HCL SERZONE E-VILL 10 SERZONE E-VILL 25 SINEQUAN SILENOR E-VILL 25 SINEQUAN SINEQUAN SEPERSOR SEPERSOR STABANIL SEFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX SUMMONTIL LAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 2-10 TETRAFON 2-25 TRIAVIL 2-25 ETRAFON 2-10 TRIAVIL 2-25 ETRAFON 4-10 TRIAVIL 2-25 ETRAFON 1-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 ETRAFON FORTE 4-25 TRIAVIL 2-7 TRIAVIL 2-8 ETRAFON FORTE 4-25 TRIAVIL 2-9 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-26 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVI | | |
| E-VILL 10 SERZONE E-VILL 100 SILENOR E-VILL 25 SINEQUAN E-VILL 50 SK-AMITRIPTYLINE E-VILL 75 SK-PRAMINE EFFEKOR STABANIL EFFEKOR STABANIL EFFEKOR XR SURMONTIL LAVIL SYMBYAX EMITIRP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNAFOR 2-10 TRIAVIL 2-10 ETRAFON 3-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 1-10 TRIAVIL 2-10 | | |
| E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR STABANIL ELAVIL SYMBYAX EMITRIP ELAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENCOPLE ENCOPL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 6-10 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON TRIAVIL 5- | | |
| SINEQUAN | | |
| E-VILL 50 E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX ELAVIL SYMBYAX ELAVIL ELAVIL ENDEP TOFRANIL-PM ENOVIL TRAZAMINE ESCITALOPRAN OXALATE ETNOFRIL ETRAFON 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-25 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-5 ETRAFON PORTE 4-25 TRIAVIL 2-5 ETRAFON PORTE 4-25 TRIAVIL 2-5 ETRAFON BORDITE 4-25 TRIAVIL 2-10 T | | |
| SK-PRAMINE | | |
| EFFEXOR STABANIL EFFEXOR XR SURMONTIL ELAVIL SYMBYAX EMITRP TOFRANIL ENDEP TOFRANIL-PM ENOVIL TRAZAMINE ENOVIL TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-5 ETRAFON 2-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 EFETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-10 FLUOX | | |
| SURMONTIL | | |
| ELAVIL SYMBYAX | | |
| EMITRIP ENDEP TOFRANIL ENDEP TOFRANILPM ENOVIL ENOVIL ENOVIL ETRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-50 FLUOVAMINE MALEATE FLUVOXAMINE FLUVOXAMINE FLUVOXAM | | |
| ENDEP FINDER FINDER FINOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-3 ETRIAVIL 2-40 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-6 ETRIAVIL 2-7 ETRIAVIL 2-8 ETRIAVIL 3-9 ETRIAVIL | | STIVIDIAX |
| ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE HCL TRIAVIL 4-50 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL 25-5 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-5 TR | I E MITDID | TOFRANII |
| TRAZODONE HCL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 FETZIMA TRIAVIL 2-7 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FORFIVO XL GABOXETINE GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL ER WANATE MIPPRAMINE HCL WINACTIL MIPRAMINE PAMOATE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 4-10 TRIAVIL 2-5 TRIAVIL 2-10 TRIAVIL 2-1 | EMITRIP | |
| ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-2 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FURD YENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL WENLAFAXINE HCL ER WANATE WIBRYD WINDERAMINE HCL WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT ZONALON | ENDEP | TOFRANIL-PM |
| ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FULOXETINE DR TRIAVIL 4-25 FULOXETINE HCL TRIAVIL 4-50 FULVOXAMINE MALEATE TRIMIPRAMINE MALEATE FULVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER IMIPRAMINE HCL VIVACTIL IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELBUTRIN JANIMINE WELBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP<br>ENOVIL | TOFRANIL-PM<br>TRAZAMINE |
| TRIAVIL 2-25 ETRAFON 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FORFIVO XL VENLAFAXINE HCL VENLAFAXINE HCL WENLAFAXINE HCL WIBRYD WIBRYD WIBRYD WIBRYD WINDERMINE HCL WINAVATE WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-5 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-2 TRIA | ENDEP ENOVIL ESCITALOPRAM OXALATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL |
| TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMPRAMINE MALEATE TRIMPRAMINE MALEATE FORFIVO XL GABOXETINE WENLAFAXINE HCL WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WELBUTRIN JANIMINE JANIMINE KENVIL KHEDEZLA ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 |
| TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE H | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 |
| TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 |
| TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 |
| FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE WENLAFAXINE HCL VENLAFAXINE HCL ER WIBRYD WIBRYD WIBRYD WIBRYD WIMIPRAMINE HCL WINACTIL WIMIPRAMINE PAMOATE WELLBUTRIN JANIMINE KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 |
| TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE ER FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIIBRYD VIIBRYD VIIBRYD VIIBRYD VIVACTIL | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 |
| FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIVACTIL MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE VELBUTRIN VELBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 |
| FORFIVO XL GABOXETINE WENLAFAXINE HCL ER WAVATE WIBRYD WIFRAMINE HCL WIFRAMINE HCL WIFRAMINE PAMOATE WELLBUTRIN WELLBUTRIN SR KENVIL KHEDEZLA KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 |
| GABOXETINE VENLAFAXINE HCL ER VIIBRYD IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELLBUTRIN IANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VONLAFAXINE HCL ER VIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE |
| MAVATE VIBRYD MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VIBRYD VIVACTIL WELLBUTRIN SR WELLBUTRIN SL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP |
| MIPRAMINE HCL MIPRAMINE PAMOATE MELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO VIVACTIL WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL |
| IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER |
| JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD |
| KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL |
| KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN |
| LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL |
| LIMBITROL ZYBAN | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON |

# Appendix A Nonbiologics

## Adalimumab

This measure categorizes the number of biologic DMARDs into the following categories:

- 0: Up to 1.0 (exclusive). This is the referent category
- 1: From 1.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 3.0 (exclusive).
- >=3: From 3.0 (inclusive) to (any)


# Certolizumab pegol


#### Etanercept


# Etanercept

| NDC Brand Name |
|------------------|
| SIMPONI |
| SIMPONI ARIA |
| NDC Generic Name |
| GOLIMUMAB |
| HCPCS |
| J1602 |

# Infliximab


# Abatacept

| NDC Brand Name |
|----------------|
| ORENCIA |


#### **Tocilizumab**


#### **Tofacitinib**

This measure categorizes the number of nonbiologic DMARDs into the following categories:

- 0: Up to 1.0 (exclusive). This is the referent category
- 1: From 1.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 2.0 (exclusive).
- 2: From 2.0 (inclusive) to 3.0 (exclusive).
- >=3: From 3.0 (inclusive) to (any)

| , |
|-----------------------------------------|
| NDC Brand Name |
| XELJANZ |
| NDC Generic Name |
| TOFACITINIB CITRATE |

#### **Auranofin**

| NDC Brand Name | | |
|------------------|-------------|---|
| RIDAURA | | |
| NDC Generic Name | | |
| AURANOFIN | | |
| NDC Drug Code | | |
| 00007487918 | 63032001160 | |
| 65483009306 | | • |

## Azathioprine

| NDC Brand Name | |
|------------------|---------------------|
| AZASAN | AZATHIOPRINE SODIUM |
| AZATHIOPRINE | IMURAN |
| NDC Generic Name | |
| AZATHIOPRINE | AZATHIOPRINE SODIUM |

# Cyclophosphamide

| NDC Brand Name | |
|------------------------------|----------------------|
| CYCLOPHOSPHAMIDE | CYTOXAN LYOPHILIZED |
| CYCLOPHOSPHAMIDE MONOHYDRATE | NEOSAR |
| CYTOXAN | NEOSAR FOR INJECTION |
| NDC Generic Name | |
| CYCLOPHOSPHAMIDE | |

#### Cyclosporine

| NDC Brand Name | |
|-----------------------|------------------------|
| CYCLOSPORINE | RESTASIS |
| CYCLOSPORINE MODIFIED | SANDIMMUNE |
| GENGRAF | SANGCYA |
| NEORAL | |
| NDC Generic Name | |
| CYCLOSPORINE | CYCLOSPORINE, MODIFIED |

# Gold sodium thiomalate

| NDC Brand Name | |
|------------------------|-------------|
| AUROLATE | MYOCHRYSINE |
| GOLD SODIUM THIOMALATE | |
| NDC Generic Name | |
| GOLD SODIUM THIOMALATE | |
| HCPCS | • |
| J1600 | |

## Leflunomide

| NDC Brand Name | |
|------------------|-------------|
| ARAVA | LEFLUNOMIDE |
| NDC Generic Name | |
| LEFLUNOMIDE | |

# Sulfasalizine

| NDC Brand Name | |
|------------------|------------------|
| AZULFIDINE | SULFASALAZINE DR |
| S.A.S500 | SULFAZINE |
| SULFA DYNE | SULFAZINE EC |
| SULFASALAZINE | |
| NDC Generic Name | |
| SULFASALAZINE | |

# Hydroxychloroquine

| NDC Brand Name | |
|------------------|------------------|
| AZULFIDINE | SULFASALAZINE DR |
| S.A.S500 | SULFAZINE |
| SULFA DYNE | SULFAZINE EC |
| SULFASALAZINE | |
| NDC Generic Name | |
| SULFASALAZINE | |

# Methotrexate

| NDC Brand Name | | |
|--------------------------------|------------------------|---|
| ABITREXATE | MEXATE | |
| FOLEX PFS | MEXATE-AQ | |
| FOLEX-PFS | OTREXUP | |
| METHOTREXATE | RASUVO | |
| METHOTREXATE LPF | RHEUMATREX | |
| METHOTREXATE SODIUM | TREXALL | |
| METHOTREXATE SODIUM PARENTERAL | | |
| NDC Generic Name | NDC Generic Name | |
| METHOTREXATE | METHOTREXATE SODIUM/PF | |
| METHOTREXATE SODIUM | METHOTREXATE/PF | |
| HCPCS | | |
| J8610 | J9260 | ` |
| J9250 | | |

# **NSAIDs and Coxibs**

| NDC Generic Name | |
|------------------|------------|
| CELECOXIB | NABUMETONE |
| DIFLUNISAL | NAPROXEN |
| ETODOLAC | OXAPROZIN |
| FLURBIPROFEN | PIROXICAM |
| IBUPROFEN | ROFECOXIB |
| INDOMETHACIN | SULINDAC |
| KETOPROFEN | VALDECOXIB |
| MELOXICAM | |

# Opioids

| Opioias | |
|--------------------------------|--------------------------|
| NDC Brand Name | |
| A-COF DH | LIQUIHISTINE CS |
| ABC COMPOUND W/CODEINE #3 | LORCET |
| ABER-TUSS HC | LORCET 10-650 |
| ABSTRAL | LORCET 10/650 |
| ACAHISTINE | LORCET HD |
| ACETA W/CODEINE | LORCET PLUS |
| ACETAMINOPH-CAFF-DIHYDROCODEIN | LORCIDE |
| ACETAMINOPHEN W-CODEINE | LORTAB |
| ACETAMINOPHEN W/CODEINE | LORTAB ASA |
| ACETAMINOPHEN-CODEINE | LORTUSS EX |
| ACTAGEN-C | LORTUSS HC |
| ACTIFED WITH CODEINE | LYNOX |
| ACTIQ | M-CLEAR |
| ADOL | M-CLEAR JR |
| AIRACOF | M-CLEAR WC |
| ALA-HIST AC | M-END |
| ALAHIST DHC | M-END MAX |
| ALCET | M-END MAX D |
| ALLAY | M-END PE |
| ALLERFRIM W/CODEINE | M-END WC |
| ALLFEN CD | M-GESIC |
| ALLFEN CDX | M-TUSS |
| ALOR | MAGNACET |
| ALPHEN | MAR-COF BP |
| AMACODONE | MAR-COF CG |
| AMAPHEN W/CODEINE NO.3 | MARCOF |
| AMBENYL | MARGESIC |
| | MARGESIC COMPOUND |
| AMBI 5/15/100 | |
| AMBIFED CD | MARGESIC H |
| AMBIFED CDX | MARGESIC IMPROVED |
| AMBIFED-G CD | MAX HC |
| AMBIFED-G CDX | MAXI-TUSS HC |
| AMBOPHEN | MAXI-TUSS HCG |
| AMGENAL | MAXI-TUSS HCX |
| AN-ABATE | MAXIDONE |
| ANACIN-3 W/CODEINE | MAXIFED CD |
| ANACIN-3 WITH CODEINE | MAXIFED CDX |
| ANAPLEX HD | MAXIFED-G CD |
| ANATUSS W/CODEINE | MAXIFED-G CDX |
| ANEXSIA | MAXIFLU CD |
| ANODYNOS-DHC | MAXIFLU CDX |
| ANOLOR DH-5 | MAXIPHEN CD |
| APOKYN | MAXIPHEN CDX |
| APOMORPHINE HCL | MAXITUSS HC |
| ASA-BUTALB-CAFFEINE-CODEINE | MC COUGH |
| ASCOMP W/CODEINE # 3 | MC JR COUGH |
| ASCOMP WITH CODEINE | MED-HIST |
| ASPIRIN W/CODEINE | MED-HIST-HC |
| ASPIRIN WITH CODEINE | MEDCODIN |
| ASPIRIN-CAFFEINE-DIHYDROCODEIN | MEDICAP HD |
| ASTRAMORPH-PF | MEDIPAIN 5 |
| ATROPINE W/DEMEROL | MEDTUSS HD |
| ATUSS EX | MEGAGESIC |
| ATUSS G | MEGAMOR |
| ATUSS HC | MEPERGAN |
| ATUSS HD | MEPERGAN FORTIS |
| ATUSS HS | MEPERIDINE HCL |
| ATUSS HX | MEPERIDINE HCL-0.9% NACL |
| ATUSS MR | MEPERIDINE HCL-NS |
| ATUSS MS | MEPERIDINE HCL-NS |
| A1000 IVID | INITE FUIDING HOLING |

| ATTUCC NIV | A A ED ED ID IN E IV /DD OA A ET IVA TIN E |
|---|---|
| ATUSS NX | MEPERIDINE W/PROMETHAZINE |
| AZDONE | MEPERIDINE-PROMETHAZINE |
| AZDONE | MEPERITAB |
| B-TUSS | MEPROZINE |
| BALACET 325 | MESEHIST WC |
| BALTUSSIN | MI-CODE |
| BALTUSSIN HC | MI-DECON |
| BANCAP HC | MINTEX HC |
| BAYCOMINE | MINTUSS EX |
| BAYCOMINE PEDIATRIC | MINTUSS G |
| BAYHISTINE | MINTUSS HC |
| BEXOPHENE | MINTUSS HD |
| BIOTUSSIN AC | MINTUSS MR |
| BIOTUSSIN DAC BIPHETANE-DC | MINTUSS MS |
| | MINTUSS NX |
| BITEX | MONTE-U LIC |
| BPM PE HC BROM-CORT-DC | MONTEFLU HC MORPHINE SULF/D5W |
| BROMANATE DC | MORPHINE SULF/NS |
| BROMANIVI | MORPHINE SULFATE |
| BROMANYL BROMAREST DC | MORPHINE SULFATE CONCENTRATE |
| BROMAREST DC | MORPHINE SULFATE CR MORPHINE SULFATE ER |
| BROMATANE-DC BROMCOMP HC | MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE |
| | MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION |
| BROMODIPHENHYDRAMINE HCL | |
| BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE | MORPHINE SULFATE O 00/ NACL |
| | MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W |
| BROMPHEN-DC | MORPHINE SULFATE/D5W MORPHINE SULFATE/D5W |
| BROMPHENEX HD BROMPHENIRAMINE DC | MORPHINE SULFATE/NS |
| DROWP HEINIKAWIINE DC | INIORPHINE SOLFATE/INS |
| | MS CONTIN |
| BROMPHENIRAMINE-DC | MS CONTIN |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE | MS/L |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE | MS/L<br>MS/S |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD | MS/L<br>MS/S<br>MSIR |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS | MS/L MS/S MSIR MULTI-HIST CS |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C | MS/L MS/S MSIR MULTI-HIST CS MYBANIL |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CB BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALBITAL COMPOUND W/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB CA BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTINAL W/CODEINE #3 C-TUSSIN | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL W/CODEINE #3 C-TUSSIN CALCIDRINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTINAL W/CODEINE #3 C-TUSSIN CALCIDRINE CALCIUM IODIDE W/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX HC BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP/CODEINE BUTINAL W/CODEINE #3 C-TUSSIN CALCIDRINE CALCIUM IODIDE W/CODEINE CANGES-HC | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NAZARIN HC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CBX BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP/CODEINE BUTINAL W/CODEINE #3 C-TUSSIN CALCIDRINE CALCIUM IODIDE W/CODEINE CANGES-HC CANGES-HC NR | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NEO AC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE C-TUSSIN CALCIDRINE CALCIUM IODIDE W/CODEINE CANGES-HC CANGES-HC NR CANGES-XP | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN AC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NEO AC NEO HC |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEIN BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL/CAFF/APAP/CODEINE CALCIDRINE CALCIDRINE CALCIUM IODIDE W/CODEINE CANGES-HC CANGES-HC CANGES-HC CANGES-XP CAPCOF | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN AC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NORCET |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CB BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE CALCIUM IODIDE W/CODEINE CALCIUM IODIDE W/CODEINE CANGES-HC CANGES-HC NR CANGES-XP CAPCOF CAPITAL W-CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN AC NALDECON-CX ADULT NALEX NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NORCET 7.5 MG |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP/CODEINE BUTALBITAL-CAFF-APAP/CODEINE BUTALBITAL-CAFF-APAP/CODEINE CALCIUM IODIDE W/CODEINE CANGES-HC CANGES-HC NR CANGES-YP CAPCOF CAPITAL W/CODEINE CAPITAL W/CODEINE CAPITAL W/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN AC NALDECON-CX ADULT NALEX NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NEO AC NOCCET NORCET 7.5 MG NORCO |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CBX BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL W/CODEINE #3 C-TUSSIN CALCIDRINE CANGES-HC CANGES-HC NR CANGES-XP CAPCOF CAPITAL W/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NORCET NORCET NORCO NOTUSS |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CB BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL COMPOUND-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL W/CODEINE #3 C-TUSSIN CALCIDRINE CANGES-HC CANGES-HC CANGES-HC CANGES-YP CAPCOF CAPITAL W/CODEINE CARISOPRODOL COMPOUND-CODEINE CARISOPRODOL COMPOUND-CODEINE CARISOPRODOL COMPOUND-CODEINE CARISOPRODOL COMPOUND-CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NORCET NORCET NORCET NORCO NOTUSS |
| BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB BROVEX CBX BROVEX CBX BROVEX PB C BROVEX PB C BROVEX PB C BROVEX PB CX BUTALB-ACETAMINOPH-CAFF-CODEIN BUTALB-CAFF-ACETAMINOPH-CODEINE BUTALBITAL COMPOUND W/CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL-CAFF-APAP-CODEINE BUTALBITAL/CAFF/APAP/CODEINE BUTALBITAL W/CODEINE #3 C-TUSSIN CALCIDRINE CANGES-HC CANGES-HC NR CANGES-XP CAPCOF CAPITAL W/CODEINE | MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE MYHYDROMINE PEDIATRIC MYPHETANE DC MYTUSSIN AC MYTUSSIN DAC NALDECON-CX ADULT NALEX NALEX AC NALEX DH NARCOF NARIZ HC NARVOX NASATUSS NASOTUSS NASOTUSS NAZARIN HC NORCET NORCET NORCEO NORCO NOTUSS |

| CGU WC | NOTUSS-FORTE |
|--------------------------------|------------------------------|
| CHEMDAL | NOTUSS-NX |
| CHEMERGAN W/CODEINE | NOTUSS-NXD |
| CHERACOL | NOTUSS-PE |
| CHERATUSSIN AC | NOVADYNE |
| CHERATUSSIN DAC | NOVADYNE DH |
| CHLORPHEN HD | NOVAGEST |
| CHLORPHENIRAMINE-CODEINE | NOVAGEST DH |
| CLEARTUSS DH | NOVAHISTINE |
| CO-GESIC | NOVAHISTINE DH |
| CO-HISTINE | NOVASUS |
| CO-HISTINE DH | NUCOCHEM |
| COASTALDYNE | NUCODINE SYR |
| COCET | NUCOFED |
| COCET PLUS | NUCOTUSS |
| CODACA NO.3 | NUDAL-HD |
| CODACA NO.4 | NUMORPHAN |
| CODAFED | OMS |
| CODAL-DH | ONCET |
| CODAMINE | ONCET 5 |
| CODAMINE PEDIATRIC | ONCET 7 |
| CODAPHEN | ONSOLIS |
| CODAR AR | OPANA |
| CODAR D | OPANA ER |
| CODAR GF | ORAMORPH SR |
| CODEFEN | ORGADIN-TUSS |
| CODEGEST | OXECTA |
| CODEINE COUGH SYRUP | OXYCODONE CONCENTRATE |
| CODEINE PHOSPHATE | OXYCODONE CONCENTRATE |
| CODEINE SULFATE | OXYCODONE HCL ER |
| CODEINE-GUAIFENESIN | OXYCODONE HCL-ACETAMINOPHEN |
| CODEINE/PHENYLPROP/GUAIFENESIN | OXYCODONE HCL-ASPIRIN |
| CODEMINE | OXYCODONE HCL-IBUPROFEN |
| CODICLEAR DH | OXYCODONE HYDROCHLORIDE |
| CODIMAL DH | OXYCODONE W/ACETAMINOPHEN |
| CODIMAL PH | OXYCODONE W/ASPIRIN |
| CODITUSS DH | OXYCODONE W/ASPIRIN HALF-STR |
| CODOTUSS | OXYCODONE-ACETAMINOPHEN |
| COLDCOUGH | OXYCODONE-ASPIRIN |
| COLDCOUGH EXP | OXYCODONE/APAP |
| COLDCOUGH HC | OXYCONTIN |
| COLDCOUGH HCM | OXYFAST |
| COLDCOUGH PD | OXYIR |
| COLDCOUGH XP | OXYMORPHONE HCL |
| COLDTUSS | OXYMORPHONE HCL ER |
| COLREX COMPOUND | P-EPD HCL/HCOD BT/CARBINOX |
| COMBUNOX | P-EPHED HCL/HYDROCOD BIT/CP |
| COMTUSSIN HC | P-TUSS |
| CONDASIN | P-TUSS D |
| CONEX W/CODEINE | P-V-TUSSIN |
| CONZIP | PALLADONE |
| COPAN | PANACET |
| COPHENE XP | PANADOL W/CODEINE NO.3 |
| COPHENE-S | PANADOL W/CODEINE NO.4 |
| CORDRON-HC | PANASAL |
| COTAB A | PANCET |
| COTAB AX | PANCOF |
| COTABFLU | PANCOF EXP |
| COTUSS EX | PANCOF HC |
| COTUSS EX | PANCOF PD |
| | PANCOF XP |
| COTUSS V | |
| COTUSS-V | PANLOR |

| [aaa=a | I |
|---|---|
| COUGHTUSS | PANLOR DC |
| CPB WC | PANLOR SS |
| CRANTEX HC | PAPA-DEINE NO.4 |
| CYCOFED | PC-CAP |
| CYNDAL | PEDIACOF |
| CYTUSS HC | PEDIATEX HC |
| CYTUSS-HC | PEDITUSS |
| D-TANN HC | PERCOCET PERCODAN |
| DAMASON-P DARVOCET A500 | PERCODAN DEMI |
| DARVOCET ASSU | PERCOLONE |
| DARVOCET-N 100 | PERLOXX |
| DARVON | PHANATUSS HC |
| DARVON COMPOUND | PHEN/CHLOR HC |
| DARVON COMPOUND 32 | PHENA-HC |
| DARVON COMPOUND-65 | PHENAPHEN W/CODEINE |
| DARVON-N | PHENDACOF HC |
| DAZIDOX | PHENDACOF PLUS |
| DE-CHLOR G | PHENERGAN VC W/CODEINE |
| DE-CHLOR HC | PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE |
| DE-CHLOR HD | PHENERGAN W/CODEINE PHENERGAN W/CODEINE |
| DE-CHLOR MR | PHENERGAN WITH CODEINE |
| DE-CHLOR NX | PHENFLU CD |
| DECOHISTINE | PHENFLU CDX |
| DECOHISTINE DH | PHENHIST |
| DECONAMINE CX | PHENYLCODONE PEDIATRIC |
| DECONGEST | PHENYLEPH-HCOD BT-CP |
| DECTUSS C | PHENYLEPHRINE HD |
| DELHISTINE CS | PHENYLHISTINE |
| DEMEROL | PHENYLHISTINE DH |
| | <del> </del> |
| DEPODUR | I PHENYLPKOP/COD/BR-PHENIKAWIINE |
| DESPEC-EXP | PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC |
| | PHENYLPROPANOLAMINE DC |
| DESPEC-EXP | |
| DESPEC-EXP<br>DESPEC-PD | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON |
| DESPEC-PD DESPEC-PDC | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHYDRO-CP | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHYDRO-CP DIHYDRO-GP | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHYDRO-CP DIHYDRO-PE | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE-BPM-PE | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-HISTINE |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST TOC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN AC POLY-TUSSIN D |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DIHYDROXCODEINE COMPOUND DIHYDROXCODEINE COMPOUND DILAUDID | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROXCODEINE COMPOUND DILAUDID DILAUDID STRIP PACKS | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN EX |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE-BPM-PE DIHYDROXCODEINE COMPOUND DILAUDID DILAUDID DILAUDID-5 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-HISTINE POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN D POLY-TUSSIN EX POLY-TUSSIN HD |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE-BPM-PE DIHYDROXCODEINE COMPOUND DILAUDID DILAUDID DILAUDID-5 DILAUDID-5 DILAUDID-1 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN AC POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-HP DIMETANE-DC | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN EX POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-HP DIMETANE-DC DOLACET | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID DILAUDID-5 DILAUDID-HP DIMETANE-DC DOLAGESIC | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-15 DILAUDID-16 DIMETANE-DC DOLAGESIC DOLENE | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-5 DILAUDID-5 DILAUDIC-5 DOLACET DOLAGESIC DOLENE DOLENE AP-65 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-HISTINE POLY-TUSSIN POLY-TUSSIN POLY-TUSSIN DD POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN CS POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-PE DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-HP DIMETANE-DC DOLACET DOLAGESIC DOLENE COMPOUND-65 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-HIST NC POLY-LSSIN POLY-HISTINE CS POLY-TUSSIN AC POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN EX POLY-TUSSIN HD POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLYGESIC POLYTINE CS POT GUAIACO-HYDROCODONE BIT PP-CAP PRIMALEV PRIMLEV |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDRO-DEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID STRIP PACKS DILAUDID-5 DILAUDID-5 DILAUDID-19 DIMETANE-DC DOLACET DOLAGESIC DOLENE COMPOUND-65 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PHURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-CS POLY-HISTINE POLY-HISTINE POLY-TUSSIN AC POLY-TUSSIN AC POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN EX POLY-TUSSIN HD POLY-TUSSIN XP |
| DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C DIHIST DH DIHISTINE DIHISTINE DIHISTINE DH DIHYDRO-CP DIHYDRO-GP DIHYDRO-PE DIHYDROCODEINE COMP MOD DIHYDROCODEINE COMPOUND DIHYDROCODEINE COMPOUND DILAUDID DILAUDID DILAUDID DILAUDID-S DILAUDID-S DILAUDID-HP DIMETANE-DC DOLACET DOLACET DOLACES DOLENE COMPOUND-65 | PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN HC POLY CS POLY HIST DHC POLY HIST DHC POLY HIST NC POLY-HIST NC POLY-LISTINE POLY-HISTINE CS POLY-TUSSIN AC POLY-TUSSIN AC POLY-TUSSIN D POLY-TUSSIN DHC POLY-TUSSIN DHC POLY-TUSSIN EX POLY-TUSSIN HD POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLY-TUSSIN XP POLYGESIC POLYTINE CS POT GUAIACO-HYDROCODONE BIT PP-CAP PRIMALEV PRIMLEV |
| DOLOREY FORTE | DDO CLEAD CADS |
|---|---|
| DOLOREX FORTE | PRO-CLEAR CAPS |
| DOLPHEN | PRO-COF D |
| DONATUSS DC DONATUSSIN DC | PRO-RED |
| DONATUSSIN MAX | PRO-RED AC |
| DORAPHEN-65 | PROCET |
| DOXAPAP N-100 | PROLEX DH |
| DRITUSS HD | PROMETHAZINE VC W/CODEINE |
| DROCON-CS | PROMETHAZINE VC-CODEINE |
| DROTUSS | PROMETHAZINE WC-CODEINE |
| DROTUSS-CP | PROMETHAZINE W/CODEINE PROMETHAZINE-CODEINE |
| DUOCET | PROPACET |
| DUOHIST DH | PROPACHEM |
| DURADAL | PROPACHEM PEDIATRIC |
| DURADAL HD | PROPAIN HC |
| DURADAL HD PLUS | PROPOXACET-N 100 |
| DURADYNE DHC | PROPOXACET-N 100 PROPOXYPHENE HCL |
| DURAGANIDIN NR | PROPOXYPHENE HCL COMPOUND |
| DURAGESIC | PROPOXYPHENE HCL W/APAP |
| DURAMORPH | PROPOXYPHENE HCL-ACETAMINOPHEN |
| DURATUSS HD | PROPOXYPHENE NCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN |
| DYNATUSS DF | PROPOXYPHENE NAPSYLATE |
| DYNATUSS HC | PROPOXYPHENE NAPSYLATE W/APAP |
| DYNATUSS HCG | PROPOXYPHENE NAPSYLATE-APAP |
| DYNEX HD | PROTEX |
| DYTAN-HC | PROTEX D |
| E-LOR | PROTUSS |
| ED TUSS HC | PROTUSS-D |
| ED-TLC | PROVAL NO.3 |
| EFASIN | PSE BPM HD |
| EFASIN | PSE BPINI HD |
| - | DCELIDATEV LIC |
| EFASIN-HD | PSEUDATEX HC |
| EFASIN-HD<br>EMBEDA | PSEUDOEPHEDRINE W/CODEINE |
| EFASIN-HD EMBEDA EMCODEINE NO.3 | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL+HD QUINTEX HC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DH | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-DH ENDACOF-HC | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-PLUS | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-PLUS ENDACOF-XP | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDAGEN-HD | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELCOF C |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDACOF-XP ENDAL | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL+DD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDACOF-XP ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN-HCX RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN RESCUDOSE |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-PLUS ENDACOF-XP ENDACOF-ND ENDAL | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN RESCUDOSE REX-A-HIST |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-PLUS ENDACOF-XP ENDACOF-ND ENDACOF-ND ENDACOF-HD ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL-HD | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDACOF-XP ENDAGEN-HD ENDAL ENDAL ENDAL ENDAL ENDAL-HD | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDACOF-XP ENDACOF-W ENDAL CD ENDAL CD ENDAL HD ENDAL HD ENDAL-HD | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELATUSS HC RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-HC ENDACOF-HC ENDACOF-AP ENDACOF-WP ENDAL ENDAL-HD ENDACOF-H ENDOCODONE | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELATUSS HC RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDAGEN-HD ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL-HD ENDOCOT E | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELATUSS HC RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-HC ENDACOF-HC ENDACOF-HC ENDACOF-WP ENDACOF-WP ENDAL HD ENDAL HD ENDAL HD ENDAL-HD ENDAL-HD ENDAL-HD PLUS ENDOCET ENDOCODONE | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELATUSS HC RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HPD |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-PLUS ENDACOF-XP ENDAGEN-HD ENDAL ENDAL ENDAL ENDAL HD ENDAL-HD ENDAL-HD ENDAL-HD PLUS ENDOCET ENDOCODONE ENDOCODONE ENDOCUSS ENPLUS-HD | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN-HCX RELATUSS HC RELATUSS HC RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HD RINDAL HPD RMS-SUPPOSITORY |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-HC ENDACOF-PLUS ENDACOF-PLUS ENDACOF-XP ENDAGEN-HD ENDAL ENDAL ENDAL CD ENDAL HD ENDAL-HD ENDAL-HD ENDAL-HD PLUS ENDOCET ENDOCODONE ENDOTUSS ENPLUS-HD ENTEX HC | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN HC RELASIN-HCX RELATUSS HC RELOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RINDAL HD RINDAL HPD RMS-SUPPOSITORY RO-CET-N 100 |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF ENDACOF-C ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-PLUS ENDACOF-PLUS ENDACOF-WP ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL ENDAL-HD END | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN HC RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD PLUS RINDAL HPD RMS-SUPPOSITORY RO-CET-N 100 ROBAFEN AC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DC ENDACOF-HC ENDACOF-HC ENDACOF-XP ENDAGEN-HD ENDAL ENDOCET ENDOCODONE E | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC RELACON-HC NR RELASIN HC RELASIN HC RELASIN HC RELATUSS HC RELOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RMS-SUPPOSITORY RO-CET-N 100 ROBAFEN AC ROBAFEN-DAC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-HC ENDACOF-XP ENDAGEN-HD ENDAL ENDAL ENDAL CD ENDAL HD ENDAL-HD ENDAL-HD ENDAL-HD PLUS ENDOCOT ENDOCOTONE ENTUSS ENPLUS-HD ENTEX HC ENTUSS ENTUSS-D ESGIC W/CODEINE | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-DD QUINTEX HC RELACON-HC RELACON-HC RELACON-HC RELASIN HC RELASIN HC RELASIN-HCX RELATUSS HC RELCOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RINDAL HD RMS-SUPPOSITORY RO-CET-N 100 ROBAFEN AC ROBAFEN-DAC ROBICHEM AC |
| EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.3 EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF AC ENDACOF-C ENDACOF-DC ENDACOF-DH ENDACOF-HC ENDACOF-YP ENDAGEN-HD ENDAL ENDOCET ENDOCODONE | PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL QUINDAL QUINDAL-HD QUINTEX HC RELACON-HC NR RELACON-HC NR RELASIN HC RELASIN HC RELASIN HC RELATUSS HC RELOF C REPREXAIN RESCUDOSE REX-A-HIST REZIRA RHINACON DH RID-A-PAIN W/CODEINE RINDAL HD RINDAL HD RINDAL HD RMS-SUPPOSITORY RO-CET-N 100 ROBAFEN AC ROBAFEN-DAC |

| EXCOF EXCOF-SF EXCLEAR EXECLEAR ROXANOL EXECLEAR-C ROXANOL SR EXECUSAR-C ROXANOL SR EXECOF-XP ROXANOL UD EXETUSS-HC ROXANOL-T EXTENDRYL HC FARBITAL W/CODEINE #3 FERRITANYL FERTANYL FENTANYL CITRATE-DSW FENTANYL CITRATE-DSW FENTANYL CITRATE-DSW FENTANYL CITRATE-SW FENTANYL CITRATE-S |
|---|
| EXECLEAR-C EXECLEAR-C ROXANOL SR EXECOF-XP ROXANOL UD EXTUSS-HC ROXANOL-T EXTENDRYL HC EXTENDRYL HC EXTENDRYL HC FARBITAL W/CODEINE #3 ROXICODONE FEERIDYNE ROXICODONE FERRIDYNE ROXICODONE FEERIDYNE ROXICODONE FERTANYL ROXIPRIN FENTANYL GITRATE FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-O.5W RYNA-C FENTANYL CITRATE-NS FENTANYL-ROPERIDOL SIMOC-HD FENTANYL-BUPIVACAINE-NS SK-65 FENTANYL-BUPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL W/TH CODEINE #3 SOMA COMPOUND W/TH CODEINE FIORINAL W/TH CODEINE #3 STAGESIC FIORINAL W/TH CODEINE STARPHEN W/CODEINE GANI-TUSS NR |
| EXECLEAR-C EXECOF-XP ROXANOL SR EXECUS-HC EXETUSS-HC ROXANOL T EXTENDRYL HC EXTENDRYL HC EXTENDRYL HC EARBITAL W/CODEINE #3 ROXICODONE FEBRIDYNE ROXICODONE FEBRIDYNE ROXICODONE FENTANYL ROXIPRIN ROXICODONE FENTANYL ROXIPRIN FENTANYL FENT |
| EXECOF-XP EXTENDRYL HC EXTENDRYL HC EARBITAL W/CODEINE #3 ROXICODONE FEBRIDYNE ROXICODONE FEBRIDYNE ROXICODONE FEBRIDYNE ROXICODONE INTENSOL FENTANYL ROXIPRIN FENTANYL BASE FENTANYL CITRATE FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL WITH DROPERIDOL SIMUC-HD FENTANYL WITH DROPERIDOL SIMUC-HD FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL BUPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYLNS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE FIORINAL W/CODEINE #3 SCAGES FIORINAL W/CODEINE #3 FIORINAL W |
| EXTENDRYL HC EXTENDRYL HC EXTENDRYL HC EXTENDRYL HC EXTENDRYL HC ERRIDIAN W/CODEINE #3 EROXICODONE FERRIDIAN W/CODEINE #3 ROXICODONE FERRIDIAN W/CODEINE #3 ROXICODONE INTENSOL FENTANYL ROXIPRIN FENTANYL FENTANYL BASE RYBIX ODT FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE-NS FENTANYL W/CODEINE FENTANYL W/DROPERIDOL SIMUC-HD FENTANYL W/THO PROPERIDOL SIMUC-HD FENTANYL W/THO PROPERIDOL SINODEINE FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTORA SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE #3 FI |
| EXTENDRYL HC FARBITAL W/CODEINE #3 ROXICODONE FEBRIDYNE ROXICODONE FEBRIDYNE ROXICODONE FERNTANYL ROXIPRIN ROXIPRIN FENTANYL BASE RYBIX ODT FENTANYL CITRATE RYDEX FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-D5W RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL OTHERE/NS S-T FORTE 2 FENTANYL WITH DROPERIDOL SIMUC-HD SIMUC-HD FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 APAP FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTORA SK-APAP W/CODEINE FENTANYL-ROPIVACINE FENTANYL-ROPIVACINE-NS FENTANYL-ROPIVACINE-NS FENTANYL-ROPIVACINE-NS FENTANYL-ROPIVACINE-NS SK-65 COMPOUND FENTANYL-ROPIVACINE-NS FENTANYL-ROPIVACINE-NS SK-65 COMPOUND FENTANYL-ROPIVACINE-NS SK-65 COMPOUND FENTANYL-ROPIVACINE-NS FENTANYL-ROPIVACINE-NS SK-65 COMPOUND FENTANYL-ROPIVACINE-NS SK-65 COMPOUND FENTANYL-ROPIVACINE-NS SK-OXYCODONE W/ASPIRIN FIORICET W/CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL W/TH CODEINE #3 SPEN-HISTINE FIORINAL W/TH CODEINE #3 SPEN-HISTINE FIORINAL W/TH CODEINE #3 SPEN-HISTINE FIORINAL W/TH CODEINE #3 SPEN-HISTINE FIORINAL W/TH CODEINE #3 STAGESIC-10 FIUTUSS NC STATUSS STARESIC-10 STATUSS STARESIC-10 STAPAYNE STOPAYNE |
| FARBITAL W/CODEINE #3 FERRIDYNE ROXICODONE INTENSOL FENTANYL ROXIPRIN FENTANYL FENTANYL BASE RYBIX ODT FENTANYL CITRATE RYDEX FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE-NS S-T FORTE 2 FENTANYL W/DROPERIDOL SIMUC-HD FENTANYL W/DROPERIDOL SINUC-HD FENTANYL-BUPIVACAINE-NS SK-65 FENTANYL-BUPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 COMPOUND FENTORA FENTANYL-SUR W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE #3 STAGESIC-10 FILUTUSS NC STERAPHEN W/CODEINE STOPAYNE FIORINS NC |
| FEBRIDYNE FENTANYL FENTANYL FENTANYL BASE FENTANYL CITRATE FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPI |
| FENTANYL BASE FENTANYL CITRATE FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL WITROPERIDOL SIMUC-HD FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL SINODEINE FENTANYL-BUPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/TH CODEINE SOMA COMPOUND W/CODEINE FIORICAL W/TH CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE F |
| FENTANYL BASE FENTANYL CITRATE RYDEX FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-DSW RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE/NS S-T FORTE 2 FENTANYL ORALET FENTANYL WITH DROPERIDOL SIMUC-HD FENTANYL WITH DROPERIDOL SINODEINE FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 APAP FENTANYL-ROPIVACAINE-NS SK-65 COMPOUND FENTORA FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORMOR W/CODEINE #3 FIORM |
| FENTANYL CITRATE FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-D5W FENTANYL CITRATE-D5W FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL ORALET FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FIORICET W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODE |
| FENTANYL CITRATE-0.9% NACL FENTANYL CITRATE-D5 W RYNA-CX FENTANYL CITRATE-NS RYZOLT FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL CITRATE/NS FENTANYL W/DROPERIDOL FENTANYL W/DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-ROPIVACAINE-NS SK-65 FENTANYL-ROPIVACAINE-NS SK-65 APAP FENTANYL/NS FENTANYL/NS FENTORA SK-APAP W/CODEINE FENTUSS FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE#3 FIORINAL W/CODEINE#5 FIORINAL W/COD |
| FENTANYL CITRATE-D5W FENTANYL CITRATE-NS FENTANYL CITRATE-NS FENTANYL CITRATE/NS FENTANYL ORALET FENTANYL W/PROPERIDOL SIMUC-HD FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTORA SK-APAP W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEI |
| FENTANYL CITRATE-NS FENTANYL CITRATE/NS S-T FORTE 2 FENTANYL WORALET SENEFEN III FENTANYL W/DROPERIDOL SIMUC-HD FENTANYL-BUPIVACAINE-NS FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS SK-65 APAP FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET W/CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND WITH CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL W/COD |
| FENTANYL CITRATE/NS FENTANYL W/DROPERIDOL FENTANYL W/TH DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL/NS FENTANYL/NS FENTANYL/NS FENTORA FENTORA FENTORA FENTORA FENTUSS FIORICET W/CODEINE FIORICET W/CODEINE FIORICET W/TODEINE FIORICET W/TODEINE FIORINAL W/CODEINE #3 FIORINAL W/TODEINE #3 FIORINAL W/CODEINE #3 FIORINAL W/ |
| FENTANYL ORALET FENTANYL W/DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL/NS FENTANYL/NS FENTORA SK-65 COMPOUND FENTUSS FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE FIORINAL W/CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE FIORINAL W/CODEI |
| FENTANYL W/DROPERIDOL FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL/ROPIVACAINE-NS FENTANYL/NS SK-65 APAP FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORMOR W/CODEINE #3 FIORMOR W/CODEINE #3 FIORMOR W/CODEINE #3 FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC-10 FLUTUSS HC STATUSS FLUTUSS AP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE STOPAYNE |
| FENTANYL WITH DROPERIDOL FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS FENTANYL/ROPIVACAINE-NS FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 FIORINAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 FIUTUSS HC STATUSS FLUTUSS XP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE STOPAYNE |
| FENTANYL-BUPIVACAINE-NS FENTANYL-ROPIVACAINE-NS SK-65 APAP FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND WITH CODEINE FIORINAL WITH CODEINE #3 SPEN-HISTINE FIORMOR W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FLUTUSS HC FLUTUSS YP STATUSS FLUTUSS YP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE STOPAYNE |
| FENTANYL-ROPIVACAINE-NS FENTANYL/NS SK-65 COMPOUND FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND WITH CODEINE FIORINAL WITH CODEINE #3 SPEN-HISTINE FIORMOR W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 FLUTUSS HC FLUTUSS YP STATUSS FLUTUSS XP STATUSS GANI-TUSS NR STOPAYNE |
| FENTANYL/NS FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORMOR W/CODEINE #3 FIORMOR W/CODEINE #3 FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 FIUTUSS HC FLUTUSS HC FLUTUSS XP STATUSS FLUTUSS XP STATUSS GREEN G-TUSS GANI-TUSS NR STOPAYNE |
| FENTORA SK-APAP W/CODEINE FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE SK-OXYCODONE W/ASPIRIN FIORICET WITH CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL WITH CODEINE #3 SPEN-HISTINE FIORMOR W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC FLUTUSS HC STATUSS FLUTUSS XP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE GANI-TUSS NR STOPAYNE |
| FENTUSS SK-OXYCODONE W/ACETAMINOPHEN FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 SOMA COMPOUND W/CODEINE FIORINAL WITH CODEINE #3 SPEN-HISTINE FIORMOR W/CODEINE #3 STAGESIC FIORTAL W/CODEINE #3 STAGESIC-10 FLUTUSS HC FLUTUSS YP STATUSS FLUTUSS XP G-TUSS STERAPHEN W/CODEINE GANI-TUSS NR STOPAYNE |
| FIORICET W/CODEINE FIORICET WITH CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIUTUSS HC FLUTUSS HC FLUTUSS XP FLUTUSS XP FLUTUSS XP FIUTUSS XP FI |
| FIORICET WITH CODEINE FIORINAL W/CODEINE #3 FIORINAL W/CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL WITH CODEINE #3 FIORINAL W/CODEINE FIORINAL W/CODEINE |
| FIORINAL W/CODEINE #3 FIORINAL WITH CODEINE #3 FIORMOR W/CODEINE #3 FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 FIUTUSS HC FLUTUSS YP G-TUSS GANI-TUSS NR SOMA COMPOUND WITH CODEINE SPEN-HISTINE STAGESIC STAGESIC-10 STAGESIC-10 STATUSS STATUSS STATUSS STATUSS GREEN STERAPHEN W/CODEINE STOPAYNE |
| FIORINAL WITH CODEINE #3 FIORMOR W/CODEINE #3 FIORTAL W/CODEINE #3 FIORTAL W/CODEINE #3 FLUTUSS HC FLUTUSS YP G-TUSS GANI-TUSS NR SPEN-HISTINE STAGESIC STAGESIC-10 STAGESIC-10 STATUSS STATUSS STATUSS STATUSS STERAPHEN W/CODEINE STOPAYNE |
| FIORMOR W/CODEINE #3 FIORTAL W/CODEINE #3 FLUTUSS HC FLUTUSS YP G-TUSS GANI-TUSS NR STAGESIC STAGESIC STAGESIC-10 STAGESIC-10 STAGESIC-10 STATUSS STATUSS STATUSS STATUSS GREEN STERAPHEN W/CODEINE STOPAYNE |
| FIORTAL W/CODEINE #3 FLUTUSS HC FLUTUSS XP STATUSS GREEN G-TUSS GANI-TUSS NR STAPHEN W/CODEINE STOPAYNE |
| FLUTUSS HC STATUSS FLUTUSS XP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE GANI-TUSS NR STOPAYNE |
| FLUTUSS XP STATUSS GREEN G-TUSS STERAPHEN W/CODEINE GANI-TUSS NR STOPAYNE |
| G-TUSS STERAPHEN W/CODEINE GANI-TUSS NR STOPAYNE |
| GANI-TUSS NR STOPAYNE |
| GECIL 100-1005 HD |
| GENAGESIC SUBLIMAZE |
| GENECOF-HC SUBSYS |
| GENECOF-XP SUDATUSS-2 GENTEX HC SUDATUSS-SF |
| GESIC-5 SUTTAR-2 |
| GESIC-HD SUTTAR-SF |
| GESTUSS-HC SYMTAN |
| GILTUSS HC SYMTAN A |
| GILTUSS PED-C SYNALGOS-DC |
| GLYDEINE SYNGESIC DC |
| GUA C SYNGESIC-DC |
| GUA PC T-GESIC |
| GUAIATUSSIN AC T-GESIC FORTE |
| GUAIFEN-C THERACODOPHEN-325 |
| GUAIFENESIN A.C. THERACODOPHEN-650 |
| GUAIFENESIN AC THERACODOPHEN-LOW-90 |
| GUAIFENESIN DAC THERATRAMADOL-60 |
| GUAIFENESIN NR THERATRAMADOL-90 |
| GUAIFENESIN W-CODEINE TL-HIST CD |
| GUAIFENESIN W/CODEINE TL-HIST CM |
| GUAIFENESIN-CODEINE TOURO HC |
| GUAIFENESIN-P-EPHEDRINE-COD TRAMADOL HCL |
| GUAIFENESIN-PHENYLEPHRINE-HCOD TRAMADOL HCL ER |
| GUAIFENESIN/CODEINE PHOSPHATE TRAMADOL HCL-ACETAMINOPHEN |
| GUAIFENESIN/P-EPHED HCL/HCOD TREZIX |

| GUAITUSSIN DAC | TRIACIN-C |
|-------------------------------|--------------------------------|
| GUAL-CO | TRIAFED WITH CODEINE |
| GUAPETEX HC | TRIAMINIC DH |
| GUIADEX DH | TRIAMINIC W/CODEINE |
| GUIAOLEX HC | TRIANT-HC |
| GUIATUSS AC | TRICODE AR |
| GUIATUSS DAC | TRICODE AR |
| GUIATUSSIN DAC | TRICODE GF TRICODENE W/CODEINE |
| GUIATUSSIN W/CODEINE | TRICOF |
| H-C TUSSIVE | TRICOF EXP |
| H-C TUSSIVE | TRICOF PD |
| HALOTUSSIN AC | TRIDAL |
| HALOTUSSIN-AC | TRIDAL HD |
| HALOTUSSIN-AC | TRIDAL HD |
| HBA | TRIFED-C |
| HC TUSSIVE-D | TRIHIST-CS |
| HC-GUAI | TRIPOSED W/CODEINE |
| HC-PE-DBROM | TRIPROLIDINE-C |
| HIST-HC | TRIPROLIDINE/P-EPHED/CODEINE |
| HIST-PLUS | TRITUSSIN |
| HISTAFED-C | TRYCET |
| HISTEX HC | TRYMINE CG |
| HISTINEX HC | TUSANA-D |
| HISTINEX PV | TUSDEC-HC |
| HISTUSS HC | TUSNEL C |
| HISTUSSIN D | TUSNEL PED-C |
| HISTUSSIN HC | TUSNEL-HC |
| НРВ МАХ | TUSS-AX |
| HPR END | TUSS-DS |
| HY-5 | TUSS-ES |
| HY-KXP | TUSS-HC |
| HY-PHEN | TUSS-PD |
| HYCET | TUSS-S |
| HYCO-PAP | TUSSADUR-HD |
| HYCODAN | TUSSAFED-HC |
| HYCODAPHEN | TUSSAFED-HCG |
| HYCOFED | TUSSAR-2 |
| HYCOGESIC | TUSSCOUGH DHC |
| HYCOMAL DH | TUSSCOUGH HC |
| HYCOMED | TUSSEND |
| HYCOMINE | TUSSHISTINE CS |
| HYCOMINE COMPOUND | TUSSI-ORGANIDIN NR |
| HYCOPHEN | TUSSI-ORGANIDIN-S NR |
| HYCOSIN | TUSSICAPS |
| НҮСОТАВ | TUSSICLEAR DH |
| HYCOTUSS | TUSSIDEN C |
| HYDEX PD | TUSSIDIN NR |
| HYDONE | TUSSIGON |
| HYDRO GP | TUSSIN AC |
| HYDRO PC II | TUSSINAL 12 |
| HYDRO PRO | TUSSINATE |
| HYDRO PRO D | TUSSIONEX |
| HYDRO-DP | TUSSIREX |
| HYDRO-PC | TUSSIVE HC |
| HYDRO-PC II PLUS | TUSSO-C |
| HYDRO-PROPANOLAMINE PEDIATRIC | TUSSO-DF |
| HYDRO-TUSS | TUSSO-HC |
| HYDRO-TUSSIN DHC | TUSSPLEX |
| HYDRO-TUSSIN EXP | TY-PAP W/CODEINE |
| HYDRO-TUSSIN HC | TY-TAB W/CODEINE |
| HYDRO-TUSSIN HD | TYLAGESIC 3 |
| HYDRO-TUSSIN HG | TYLENOL W/CODEINE |
| | <del>-</del> |

| LIVERO TUCCIN VE | TVI FNOL IN/CODEINE NO 2 |
|---|---|
| HYDRO-TUSSIN XP | TYLENOL W/CODEINE NO.2 |
| HYDROCOT HYDROCOD BIT-PHENYLEPHRINE-CP | TYLENOL W/CODEINE NO.4 |
| HYDROCOD-CPM-PSEUDOEPHEDRINE | TYLENOL W/CODEINE NO.4 TYLENOL-CODEINE NO.3 |
| HYDROCOD/CARBINOX/PSEUDOEPHED | TYLENOL-CODEINE NO.4 |
| HYDROCODONE | TYLOX |
| HYDROCODONE BIT-HOMATROPINE MB | UGESIC |
| HYDROCODONE BIT-HOMATKOPINE IVIB | ULTRACET |
| HYDROCODONE BIT-IBOTROTEN HYDROCODONE BITARTRATE | ULTRAGESIC |
| HYDROCODONE BT-HOMATROPINE MBR | ULTRAM |
| HYDROCODONE COMPOUND | ULTRAM ER |
| HYDROCODONE CP | UMI-APAP |
| HYDROCODONE GF | UNI MULTIHIST CS |
| HYDROCODONE HD | UNITUSS HC |
| HYDROCODONE PA | UNI-COF |
| HYDROCODONE W-ACETAMINOPHEN | UNI-COF EXP |
| HYDROCODONE W/ACETAMINOPHEN | UNI-LEV |
| HYDROCODONE W/GUAIFENESIN | UNI-TRICOF HC |
| HYDROCODONE W/PHENYLPROP | VANACET |
| HYDROCODONE-ACETAMINOPHEN | VANACOF CD |
| HYDROCODONE-GUAIFENESIN | VANACON |
| HYDROCODONE-HOMATROPINE | VANEX GRAPE |
| HYDROCODONE-HOMATROPINE MBR | VANEX HD |
| HYDROCODONE-IBUPROFEN | VAZOTUSS HC |
| HYDROCODONE-POT GUAIACOSULFON | VENDONE |
| HYDROCODONE/ACETAMINOPHEN | VERDROCET |
| HYDROCODONE/HOMATROPINE | VI-Q-TUSS |
| HYDROCODONE/PHENYLEPH/PYRILAM | VICOCLEAR DH |
| HYDROCODONE/PHENYLPROPANOLAMIN | VICODIN |
| HYDROCOF-HC | VICODIN ES |
| HYDROFED | VICODIN HP |
| HYDROGESIC | VICODIN TUSS |
| HYDROMET | VICOPROFEN |
| HYDROMET<br>HYDROMINE | VICOPROFEN VIHISTINE |
| HYDROMINE | VIHISTINE |
| HYDROMINE<br>HYDROMINE PEDIATRIC | VIHISTINE<br>VIRTUSSIN AC |
| HYDROMINE HYDROMINE PEDIATRIC HYDROMORPHONE ER | VIHISTINE VIRTUSSIN AC VISVEX HC |
| HYDROMINE HYDROMINE PEDIATRIC HYDROMORPHONE ER HYDROMORPHONE HCL | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE |
| HYDROMINE HYDROMINE PEDIATRIC HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN |
| HYDROMINE HYDROMINE PEDIATRIC HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC XARTEMIS XR |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON KGS HYDRON PSC | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 5-300 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPANE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 5-300 XODOL 7.5-300 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPANE HYDROPHEN | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 5-300 XODOL 7.5-300 XOLOX |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON CP HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON CP HYDRON KGS HYDRON FSC HYDROPHEN HYDROPHEN HYDROPHEN | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS EXP WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON CP HYDRON KGS HYDRON PSC HYDROPANE HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHENE DH HYDROPHENE DH HYDROPHENE DH | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10-300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON KGS HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN PEDIATRIC HYDROSTAT HYPHED | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC Z-COF HC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON KGS HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN PEDIATRIC HYDROPHENE DH HYDROSTAT HYPHED HYPHEN-HD | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC Z-COF HCX Z-TUSS 2 |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL-NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPANE HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROSTAT HYPHED HYPHEN-HD HYTAN | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 7.5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC Z-COF HC Z-TUSS 2 Z-TUSS AC |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON KGS HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN HYDROSTAT HYPHED HYPHEN-HD HYTAN IBUDONE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC Z-COF HC Z-TUSS E |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN PEDIATRIC HYDROPHENE DH HYDROSTAT HYPHED HYPHEN-HD HYTAN IBUDONE IDENAL W/CODEINE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10-300 XODOL 5-300 XODOL 5-300 XODOL 7.5-300 XODOL 7.5-300 XOPOCT-HC XYLON 10 Z-COF HC Z-COF HCX Z-TUSS 2 Z-TUSS E ZAMICET |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPHENE HYDROPHENE HYDROPHENE HYDROPHENE HYDROPHENE DH HYDROPHENE DH HYDROSTAT HYPHED HYPHEN-HD HYTAN IBUDONE IDENAL W/CODEINE INFUMORPH | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10/300 XODOL 5-300 XODOL 5-300 XODOL 7.5-300 XOLOX XPECT-HC XYLON 10 Z-COF HC Z-COF HC Z-TUSS AC Z-TUSS E ZAMICET ZERLOR |
| HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL HYDROMORPHONE HCL HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W HYDROMORPHONE HCL-NS HYDROMORPHONE HCL/NS HYDROMORPHONE HYDROCHLORIDE HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS HYDROMORPHONE/BUPIVACAINE HYDROMORPHONE/BUPIVACAINE HYDRON CP HYDRON EX HYDRON KGS HYDRON PSC HYDROPHEN HYDROPHEN HYDROPHEN HYDROPHEN PEDIATRIC HYDROPHENE DH HYDROSTAT HYPHED HYPHEN-HD HYTAN IBUDONE IDENAL W/CODEINE | VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ VOPAC W/W-HISTINE WELL-TUSS HD WELLTUSS HC WYGESIC XARTEMIS XR XODOL 10-300 XODOL 10-300 XODOL 5-300 XODOL 5-300 XODOL 7.5-300 XODOL 7.5-300 XOPOCT-HC XYLON 10 Z-COF HC Z-COF HCX Z-TUSS 2 Z-TUSS E ZAMICET |

| [10.551.0.15 | 707774 4000 |
|---|---|
| IOFEN-C NF | ZODRYL AC 30 |
| IOPHEN | ZODRYL AC 35 |
| IOPHEN C-NR | ZODRYL AC 40 |
| IOPHEN-C NR | ZODRYL AC 50 |
| IOTUSSIN D | ZODRYL AC 60 |
| IOTUSSIN HC | ZODRYL AC 80 |
| ISOBUTAL W/CODEINE | ZODRYL DAC 25 |
| ISOLIN W/CODEINE | ZODRYL DAC 30 |
| ISOLLYL W/CODEINE | ZODRYL DAC 35 |
| J-CET | ZODRYL DAC 40 |
| J-COF DHC | ZODRYL DAC 50 |
| J-MAX DHC | ZODRYL DAC 60 |
| J-TAN D HC | ZODRYL DAC 80 |
| JAYCOF LIC | ZODRYL DEC 25 |
| JAYCOF-HC | ZODRYL DEC 30 |
| JAYCOF-XP | ZODRYL DEC 35 |
| KADIAN | ZODRYL DEC 40 |
| KG-DAL HD | ZODRYL DEC 50 |
| KG-DAL HD PLUS | ZODRYL DEC 80 |
| KG-FED | ZODRYL DEC 80 |
| KG-FED PEDIATRIC | ZOLYIT |
| KG-TUSS HD | ZOLVIT |
| KG-TUSSIN | ZOTEX LIC |
| KGS-HC | ZOTEX-HC |
| KWELCOF | ZTUSS THE STATE OF |
| LAZANDA | ZTUSS ZT |
| LEVALL | ZUTRIPRO |
| LEVALL 5.0 | ZYDONE |
| LEXUSS 210 | ZYMINE HC |
| LIQUICET | ZYRPHEN-HC |
| LIQUICOUGH HC | |
| NDC Generic Name | WEDEDIDINE HOLIN O 0 % SODILIM CHI ODIDE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MEPERIDINE HCL IN 0.9 % SODIUM CHLORIDE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5 % WATER/PF |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE/ASPIRIN |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE SULFATE CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE SULFATE CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE SULFATE CODEINE/SSPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE/SAPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE II DOSOMAL/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE/SAPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE/POTASSIUM |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE SULFATE CODEINE/SAPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE SULFATE CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE SULFATE CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/GUAIFENESIN DIHYDROCODEINE/ASPIRIN/CAFFEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/DIHYDROCODEINE BITARTRATE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE/SAPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/GUAIFENESIN DIHYDROCODEINE/ASPIRIN/CAFFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE DIPHENHYDRAMINE HCL/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/DEXTROSE 5% WATER/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/DIHYDROCODEINE PHENYLEPHRINE HCL/DIHYDROCODEINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/GUAIFENESIN DIHYDROCODEINE BITARTRATE/GUAIFENESIN DIHYDROCODEINE/ASPIRIN/CAFFEINE DIPHENHYDRAMINE HCL/PHENYLEPHRINE HCL/CODEINE FENTANYL | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/NALTREXONE HCL MORPHINE SULFATE/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/DIHYDROCODEINE PHENYLEPHRINE HCL/DIHYDROCODEINE PHENYLEPHRINE HCL/DIHYDROCODEINE PHENYLEPHRINE HCL/DIHYDROCODEINE |
| NDC Generic Name BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE BROMPHENIRAMINE MALEATE/PHENYLEPHRINE BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE CHLORPHENIRAMINE MALEATE/CODEINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE CODEINE PHOSPHATE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE PHOSPHATE/PYRILAMINE MALEATE CODEINE/SAPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE CODEINE/CALCIUM IODIDE DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIHYDROCODEINE BITARTRATE/GUAIFENESIN DIHYDROCODEINE/ASPIRIN/CAFFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE DIPHENHYDRAMINE HCL/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF MEPERIDINE HCL/PROMETHAZINE HCL MORPHINE SULFATE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE/PF MORPHINE SULFATE LIPOSOMAL/PF MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF MORPHINE SULFATE/DEXTROSE 5% WATER/PF OXYCODONE HCL OXYCODONE HCL OXYCODONE HCL/ACETAMINOPHEN OXYCODONE HCL/ASPIRIN OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN OXYCODONE/ASPIRIN OXYMORPHONE HCL PHENYLEPHRINE HCL/CODEINE PHOSPHATE PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN PHENYLEPHRINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/CODEINE/PYRILAMINE PHENYLEPHRINE HCL/DIHYDROCODEINE PHENYLEPHRINE HCL/DIHYDROCODEINE |

# Appendix A Nonbiologics

| FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM | PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES |
|---|---|
| FENTANYL CITRATE/DEXTROSE 5% WATER/PF | PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE |
| FENTANYL CITRATE/DROPERIDOL | PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE |
| FENTANYL CITRATE/PF | POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE |
| FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF | PROMETHAZINE HCL/CODEINE |
| GUAIFENESIN/CODEINE PHOSPHATE | PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE |
| GUAIFENESIN/HYDROCODONE BITARTRATE | PROPOXYPHENE HCL |
| GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE | PROPOXYPHENE HCL/ACETAMINOPHEN |
| GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| GUAIFENESIN/PHENYLPROPANOLAMINE | PROPOXYPHENE NAPSYLATE |
| GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE | PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN |
| GUAIFENESIN/PSEUDOEPHEDRINE | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE |
| HYDROCODONE BITARTRATE | PSEUDOEPHEDRINE HCL/CODEINE |
| HYDROCODONE BITARTRATE/ACETAMINOPHEN | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE |
| HYDROCODONE BITARTRATE/ASPIRIN | PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE |
| HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE | PSEUDOEPHEDRINE HCL/DIHYDROCODEINE |
| HYDROCODONE BITARTRATE/HOMATROPINE METHYLBROMIDE | PSEUDOEPHEDRINE HCL/HYDROCODONE BITARTRATE |
| HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE | PSEUDOEPHEDRINE HCL/HYDROCODONE |
| HYDROCODONE/IBUPROFEN | PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE |
| HYDROMORPHONE HCL | PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE |
| HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE | PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE |
| HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF | PYRILAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE PHOSPHATE |
| HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF | PYRILAMINE MALEATE/PHENYLEPHRINE HCL/DIHYDROCODEINE BT |
| HYDROMORPHONE HCL/BUPIVACAINE HCL IN 0.9% SODIUM | PYRILAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE |
| HYDROMORPHONE HCL/PF | TRAMADOL HCL |
| IBUPROFEN/OXYCODONE HCL | TRAMADOL HCL/ACETAMINOPHEN |
| MEPERIDINE HCL | |

### Glucocorticoids

| Ingredient code | |
|---------------------------|----------------------|
| P5AR - prednisone | P5BC - dexamethasone |
| P5CB - triamcinolone | P5BB - betamethasone |
| P5AM - methylprednisolone | P5BL - budesonide |
| P5AB - hydrocortisone | P5AH - prednisolone |
| P5AA - cortisone | |

## Appendix A Comorbid conditions

**Atrial Fibrillation** 


Heart Failure


Stroke or TIA


| 163312 43401 163313 43401 163321 43401 163322 43401 163323 43401 163329 43401 163331 163331 43401 163331 163331 | Cerebral infarction due to thrombosis of left middle cerebral artery Cerebral infarction due to thrombosis of bilateral middle cerebral arteries Cerebral infarction due to thrombosis of unspecified middle cerebral artery Cerebral infarction due to thrombosis of right anterior cerebral artery Cerebral infarction due to thrombosis of left anterior cerebral artery Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior cerebral artery | Cerebral thrombosis with cerebral infarction |
|---|---|---|
| 163319 43401<br> 163321 43401<br> 163322 43401<br> 163323 43401<br> 163329 43401<br> 163331 43401 | Cerebral infarction due to thrombosis of bilateral middle cerebral arteries Cerebral infarction due to thrombosis of unspecified middle cerebral artery Cerebral infarction due to thrombosis of right anterior cerebral artery Cerebral infarction due to thrombosis of left anterior cerebral artery Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior | Cerebral thrombosis with cerebral infarction Cerebral thrombosis with cerebral infarction Cerebral thrombosis with cerebral infarction |
| 163321 | Cerebral infarction due to thrombosis of unspecified middle cerebral artery Cerebral infarction due to thrombosis of right anterior cerebral artery Cerebral infarction due to thrombosis of left anterior cerebral artery Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior | Cerebral thrombosis with cerebral infarction Cerebral thrombosis with cerebral infarction |
| 163322 | Cerebral infarction due to thrombosis of right anterior cerebral artery Cerebral infarction due to thrombosis of left anterior cerebral artery Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior | Cerebral thrombosis with cerebral infarction |
| 163323 43401<br>163329 43401<br>163331 43401 | Cerebral infarction due to thrombosis of left anterior cerebral artery Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior | |
| I63329 43401<br>I63331 43401 | Cerebral infarction due to thrombosis of bilateral anterior arteries Cerebral infarction due to thrombosis of unspecified anterior | Cerebral thrombosis with cerebral infarction |
| l63331 43401 | Cerebral infarction due to thrombosis of unspecified anterior | |
| | cerebral artery | Cerebral thrombosis with cerebral infarction |
| | Cerebral infarction due to thrombosis of right posterior | Cerebral thrombosis with cerebral infarction |
| 163332 43401 | Cerebral infarction due to thrombosis of left posterior | Cerebral thrombosis with cerebral infarction |
| 163333 43401 | cerebral artery Cerebral infarction to thrombosis of bilateral posterior | Cerebral thrombosis with cerebral infarction |
| 163339 43401 | Cerebral infarction due to thrombosis of unspecified posterior | Cerebral thrombosis with cerebral infarction |
| l63341 43401 | Cerebral infarction due to thrombosis of right cerebellar | Cerebral thrombosis with cerebral infarction |
| 163342 43401 | Cerebral infarction due to thrombosis of left cerebellar | Cerebral thrombosis with cerebral infarction |
| 163343 43401 | Cerebral infarction to thrombosis of bilateral cerebellar | Cerebral thrombosis with cerebral infarction |
| 163349 43401 | Cerebral infarction due to thrombosis of unspecified | Cerebral thrombosis with cerebral infarction |
| 16339 43401 | Cerebral infarction due to thrombosis of other cerebral | Cerebral thrombosis with cerebral infarction |
| 1636 43401 | Cerebral infarction due to cerebral venous thrombosis, | Cerebral thrombosis with cerebral infarction |
| I6340 43411 | Cerebral infarction due to embolism of unspecified cerebral artery | Cerebral embolism with cerebral infarction |
| l63411 43411 | Cerebral infarction due to embolism of right middle cerebral artery | Cerebral embolism with cerebral infarction |
| l63412 43411 | Cerebral infarction due to embolism of left middle cerebral artery | Cerebral embolism with cerebral infarction |
| 163413 43411 | Cerebral infarction due to embolism of bilateral middle cerebral arteries | Cerebral embolism with cerebral infarction |
| l63419 43411 | Cerebral infarction due to embolism of unspecified middle cerebral artery | Cerebral embolism with cerebral infarction |
| l63421 43411 | Cerebral infarction due to embolism of right anterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163422 43411 | Cerebral infarction due to embolism of left anterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163423 43411 | Cerebral infarction due to embolism of bilateral anterior cerebral arteries | Cerebral embolism with cerebral infarction |
| 163429 43411 | Cerebral infarction due to embolism of unspecified anterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163431 43411 | Cerebral infarction due to embolism of right posterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163432 43411 | Cerebral infarction due to embolism of left posterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163433 43411 | Cerebral infarction due to embolism of bilateral posterior cerebral arteries | Cerebral embolism with cerebral infarction |
| 163439 43411 | Cerebral infarction due to embolism of unspecified posterior cerebral artery | Cerebral embolism with cerebral infarction |
| 163441 43411 | Cerebral infarction due to embolism of right cerebellar artery | Cerebral embolism with cerebral infarction |


## Peripheral vascular disease


| Unspecified atherosclerosis of other type of bypass graft(s) of the extremities, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, right leg 170712 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, left leg 170713 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, bilateral legs 170718 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, bilateral legs 170719 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity 170721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170731 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity |
|---|
| 170711 |
| extremities with intermittent claudication, right leg 170712 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, left leg 170713 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, bilateral legs 170718 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, other extremity 170719 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity 170721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, left leg 170713 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, bilateral legs 170718 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, other extremity 170719 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity 170721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with intermittent claudication, left leg 170713 |
| Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, bilateral legs Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, other extremity Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the restremity |
| extremities with intermittent claudication, bilateral legs Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, other extremity Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| I70718 |
| extremities with intermittent claudication, other extremity 170719 Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity 170721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| Atherosclerosis of other type of bypass graft(s) of the extremities with intermittent claudication, unspecified extremity I70721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg I70722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg I70723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs I70728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity I70729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity I70731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with intermittent claudication, unspecified extremity 170721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| I70721 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, right leg I70722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg I70723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs I70728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity I70729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity I70731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with rest pain, right leg 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| 170722 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with rest pain, left leg 170723 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, bilateral legs 170728 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with rest pain, bilateral legs Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity Atherosclerosis of other type of bypass graft(s) of the right |
| Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with rest pain, other extremity 170729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| I70729 Atherosclerosis of other type of bypass graft(s) of the extremities with rest pain, unspecified extremity I70731 Atherosclerosis of other type of bypass graft(s) of the right |
| extremities with rest pain, unspecified extremity 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| 170731 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of thigh |
| 170732 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of calf |
| 170733 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of ankle |
| 170734 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of heel and midfoot |
| 170735 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of other part of foot |
| 170738 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of other part of lower leg |
| 170739 Atherosclerosis of other type of bypass graft(s) of the right |
| leg with ulceration of unspecified site |
| 170741 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of thigh |
| 170742 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of calf |
| 170743 Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of ankle |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of heel and midfoot Atheresolaters is of other type of hypers graft(s) of the left leg |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of other part of foot |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of other part of lower leg |
| Atherosclerosis of other type of bypass graft(s) of the left leg |
| with ulceration of unspecified site |
| Atherosclerosis of other type of bypass graft(s) of other |
| extremity with ulceration |
| Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, right leg |
| 170762 Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, left leg |
| 170763 Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, bilateral legs |
| 170768 Atherosclerosis of other type of bypass graft(s) of the |
| extremities with gangrene, other extremity |

# Appendix A Comorbid conditions


Hyperlipidemia

| Hypernplaci | туретпристи | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
| E780 | 2720 | Pure hypercholesterolemia | PURE HYPERCHOLESTEROLEMIA |
| E7800 | 2722 | | MIXED HYPERLIPIDEMIA |
| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED PATHOLOGICA |
|---|---|---|---|
| | | mesangiocapillary glomerulonephritis | LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense deposit disease | CHRONIC GLOMERULONEPHRITIS WITH LESION OF PROLIFERATIVE GLOMERULONEPHRITIS |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | CHRONIC GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | morphologic changes | PROGRESSIVE GLOMERULONEPHRITIS |
| N020 | 5828 | Recurrent and persistent hematuria with minor glomerular | CHRONIC GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| | | abnormality | PATHOLOGICAL LESION IN KIDNEY |
| N021 | 5829 | Recurrent and persistent hematuria with focal and | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED |
| | | segmental glomerular lesions | PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| - | | membranous glomerulonephritis | OR CHRONIC WITH LESION OF PROLIFERATIVE |
| | | Section 2 Sectio | GLOMERULONEPHRITIS |
| N023 | 5831 | Recurrent and persistent hematuria with diffuse mesangial | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | 5552 | proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOUS |
| | | promerative gromeratoric printers | GLOMERULONEPHRITIS |
| N024 | 5832 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| 11024 | 3632 | endocapillary proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOPROLIFERATIVE |
| | | endocapinary promerative giorner dionephiritis | GLOMERULONEPHRITIS |
| NOOF | F024 | Description of requirement because with differen | |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | mesangiocapillary glomerulonephritis | OR CHRONIC WITH LESION OF RAPIDLY PROGRESSIVE |
| | | | GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | disease | OR CHRONIC WITH LESION OF RENAL CORTICAL NECROSIS |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse crescentic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | glomerulonephritis | OR CHRONIC WITH LESION OF RENAL MEDULLARY NECROSI |
| N028 | 5838 | Recurrent and persistent hematuria with other morphologic | |
| | | changes | OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESIC |
| | | | IN KIDNEY |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified | |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| N029 | 5839 | _ <b> </b> | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| N029<br>N030 | 5839<br>5846 | _ <b> </b> | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN<br>KIDNEY |
| | | morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN<br>KIDNEY |
| | | morphologic changes Chronic nephritic syndrome with minor glomerular | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS |
| N030 | 5846 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE<br>OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN<br>KIDNEY<br>ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL |
| N030 | 5846 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA |
| N030<br>N031 | 5846<br>5847 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS |
| N030<br>N031 | 5846<br>5847 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED |
| N030<br>N031<br>N032 | 5846<br>5847<br>5848 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N030<br>N031<br>N032 | 5846<br>5847<br>5848 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N030<br>N031<br>N032<br>N033 | 5846<br>5847<br>5848<br>5849 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED |
| N030<br>N031<br>N032<br>N033<br>N034 | 5846<br>5847<br>5848<br>5849<br>5851 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE I |
| N030<br>N031<br>N032<br>N033 | 5846<br>5847<br>5848<br>5849 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED |
| N030<br>N031<br>N032<br>N033<br>N034 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE I |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N030<br>N031<br>N032<br>N033<br>N034 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease Chronic nephritic syndrome with diffuse crescentic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE I |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease Chronic nephritic syndrome with diffuse crescentic glomerulonephritis | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE I CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854<br>5855 | Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease Chronic nephritic syndrome with diffuse crescentic glomerulonephritis Chronic nephritic syndrome with other morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854<br>5855 | Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with diffuse crescentic glomerulonephritis Chronic nephritic syndrome with other morphologic changes Chronic nephritic syndrome with other morphologic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICA NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULD (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037<br>N038 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854<br>5855<br>5856 | Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with diffuse crescentic glomerulonephritis Chronic nephritic syndrome with other morphologic changes Chronic nephritic syndrome with other morphologic changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) CHRONIC KIDNEY DISEASE STAGE V END STAGE RENAL DISEASE CHRONIC KIDNEY DISEASE |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037<br>N038<br>N039 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854<br>5855<br>5856<br>5859 | morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease Chronic nephritic syndrome with diffuse crescentic glomerulonephritis Chronic nephritic syndrome with other morphologic changes Chronic nephritic syndrome with unspecified morphologic changes Nephrotic syndrome with minor glomerular abnormality | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) CHRONIC KIDNEY DISEASE STAGE V END STAGE RENAL DISEASE CHRONIC KIDNEY DISEASE UNSPECIFIED UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND |
| N030<br>N031<br>N032<br>N033<br>N034<br>N035<br>N036<br>N037<br>N038<br>N039 | 5846<br>5847<br>5848<br>5849<br>5851<br>5852<br>5853<br>5854<br>5855<br>5856<br>5859 | Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary proliferative glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with diffuse mesangiocapillary glomerulonephritis Chronic nephritic syndrome with dense deposit disease Chronic nephritic syndrome with diffuse crescentic glomerulonephritis Chronic nephritic syndrome with other morphologic changes Chronic nephritic syndrome with unspecified morphologic changes Nephrotic syndrome with minor glomerular abnormality | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED CHRONIC KIDNEY DISEASE STAGE II (MILD) CHRONIC KIDNEY DISEASE STAGE III (MODERATE) CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) CHRONIC KIDNEY DISEASE STAGE V END STAGE RENAL DISEASE |

| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative | INJURY TO KIDNEY WITH OPEN WOUND INTO CAVITY |
|---|---|---|---|
| N044 | | glomerulonephritis Nephrotic syndrome with diffuse endocapillary proliferative | |
| | | glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic | |
| N048 | | glomerulonephritis Nephrotic syndrome with other morphologic changes | |
| N048 | | Nephrotic syndrome with other morphologic changes Nephrotic syndrome with unspecified morphologic changes | |
| N050 | | Unspecified nephritic syndrome with minor glomerular | |
| | | abnormality | |
| N051 | | Unspecified nephritic syndrome with focal and segmental glomerular lesions | |
| N052 | | Unspecified nephritic syndrome with diffuse membranous glomerulonephritis | |
| N053 | | Unspecified nephritic syndrome with diffuse mesangial proliferative glomerulonephritis | |
| N054 | | Unspecified nephritic syndrome with diffuse endocapillary | |
| | | proliferative glomerulonephritis | |
| N055 | | Unspecified nephritic syndrome with diffuse | |
| | | mesangiocapillary glomerulonephritis | |
| N056 | | Unspecified nephritic syndrome with dense deposit disease | |
| N057 | | Unspecified nephritic syndrome with diffuse crescentic | |
| | | glomerulonephritis | |
| N058 | | Unspecified nephritic syndrome with other morphologic changes | |
| N059 | | Unspecified nephritic syndrome with unspecified | |
| 14055 | | morphologic changes | |
| N060 | | Isolated proteinuria with minor glomerular abnormality | |
| N061 | | Isolated proteinuria with focal and segmental glomerular | |
| | | lesions | |
| N062 | | Isolated proteinuria with diffuse membranous | |
| | | glomerulonephritis | |
| N063 | | Isolated proteinuria with diffuse mesangial proliferative | |
| N064 | | glomerulonephritis | |
| NU04 | | Isolated proteinuria with diffuse endocapillary proliferative glomerulonephritis | |
| N065 | | Isolated proteinuria with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N066 | | Isolated proteinuria with dense deposit disease | |
| N067 | | Isolated proteinuria with diffuse crescentic | |
| | | glomerulonephritis | |
| N068 | | Isolated proteinuria with other morphologic lesion | |
| N069 | | Isolated proteinuria with unspecified morphologic lesion | |
| N070 | | Hereditary nephropathy, not elsewhere classified with | |
| NO71 | | minor glomerular abnormality | |
| N071 | | Hereditary nephropathy, not elsewhere classified with focal and segmental glomerular lesions | |
| N072 | | Hereditary nephropathy, not elsewhere classified with | |
| | | diffuse membranous glomerulonephritis | |
| N073 | | Hereditary nephropathy, not elsewhere classified with | |
| | | diffuse mesangial proliferative glomerulonephritis | |
| N074 | | Hereditary nephropathy, not elsewhere classified with | |
| NOZE | | diffuse endocapillary proliferative glomerulonephritis | |
| N075 | | Hereditary nephropathy, not elsewhere classified with diffuse mesangiocapillary glomerulonephritis | |
| N076 | | Hereditary nephropathy, not elsewhere classified with | |
| | | dense deposit disease | |
| N077 | | Hereditary nephropathy, not elsewhere classified with | |
| | | diffuse crescentic glomerulonephritis | |


Chronic liver disease


### Asthma

